**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301

Version: 3.0 / 31Jan2023

## **Clinical Study Protocol**

A MULTICENTER, PROSPECTIVE, RANDOMIZED, CONTROLLED, OPEN LABEL TRIAL TO EVALUATE THE SAFETY AND EFFICACY OF MYNX CONTROL™ VENOUS VASCULAR CLOSURE DEVICE 6F-12F VS. MANUAL COMPRESSION IN PATIENTS WHO HAVE UNDERGONE ENDOVASCULAR PROCEDURES UTILIZING UP TO 12F PROCEDURAL SHEATHS ReliaSeal

Protocol Number: P22-8301
Cordis Document Control Number: 100606833
Protocol Version/Date: 3.0 / 31Jan2023

Product: MYNX CONTROL™ Venous Vascular Closure Device 6F-12F

Model/Specification: MX61260

Sponsor's Name/Address: Cordis US Corp.
14201 NW 60<sup>th</sup> Ave

Miami Lakes, FL 33014

Javier Sanchez, MD

National Principal Investigator

Name/Address:

Medical City Dallas Heart Hospital 11970 North Central Expressway

Dallas, TX 75243

Registration Number(s): NCT005554471

Author Name: Jenny Jimenez, Sr Clinical Project Manager

#### **Version History**

| Version Number | Version Date | Summary of Revisions |
|---|---|---|
| 1.0 | 25May2022 | N/A (original version) |
| 1.1 | 27May2022 | Administrative Changes. |
| 2.0 | 13Nov2022 | Changes to address FDA's study design considerations and clarifications for Investigational sites |
| 3.0 | 31Jan2023 | Addresses FDA's considerations from the 19Jan2023 letter |

The information in this document is the property of Cordis and is CONFIDENTIAL and PROPRIETARY. Neither the document nor the information contained therein may be reproduced or disclosed outside Cordis without the written consent of the company.




100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


A MULTICENTER, PROSPECTIVE, RANDOMIZED, CONTROLLED, OPEN LABEL TRIAL TO EVALUATE THE SAFETY AND EFFICACY OF MYNX CONTROL™ VENOUS VASCULAR CLOSURE DEVICE 6F12F VS. MANUAL COMPRESSION IN PATIENTS WHO HAVE UNDERGONE ENDOVASCULAR
PROCEDURES UTILIZING UP TO 12F PROCEDURAL SHEATHS

ReliaSeal Protocol Number: P22-8301 Version: 3.0 Version Date: 31Jan2023

#### **Approval Signatures**

# I AM THE PRIMARY AUTHOR OF THIS STUDY PROTOCOL AND CONFIRM TO THE BEST OF MY KNOWLEDGE IT IS COMPLETE AND ACCURATE.

| Name | Role | Signature | Date |
|---|---|---|---|
| Jenny Jimenez | Clinical Project Manager | //ENNY //MENE// Reason | nically signed by: Jenny Jimenez<br>: Reviewed<br>eb 3, 2023 09:54 EST |

# I HAVE REVIEWED THE STUDY PROTOCOL AND CONFIRM TO THE BEST OF MY KNOWLEDGE IT IS COMPLETE AND ACCURATE.

| Name | Role | Signature | Date |
|---|---|---|---|
| Dr. Nusrath Sultana | Medical Monitor | Electroni<br>Reason:<br>Date: Fel | pally signed by: Nusrath Sultana<br>Approved<br>3, 2023 07:03 PST |
| Steve Ullery | Statistician | Steven Ullery Reason. | ically signed by: Steven Ullery<br>Reviewed<br>b 3, 2023 09:54 PST |
| Crystal Placona | Regulatory Affairs | Crystal Placona Reason:<br>Date: Fe | dally signed by: Crystal Placona<br>Approved<br>53, 2023 10:02 EST |
| Dr Nusrath Sultana | Clinical Management | Reason: | ically signed by: Nusrath Sultana<br>Approved<br>3, 2023 07:03 PST |

| | | |
|--------------|--------------|-------------|

Protocol Clinical Clinical Study

Evaluation of Safety and Efficacy of Mynx Control Venous Vascular Closure Device 6F-12F (ReliaSeal)

Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


A MULTICENTER, PROSPECTIVE, RANDOMIZED, CONTROLLED, OPEN LABEL TRIAL TO EVALUATE THE SAFETY AND EFFICACY OF MYNX CONTROL™ VENOUS VASCULAR CLOSURE DEVICE 6F-12F VS. MANUAL COMPRESSION IN PATIENTS WHO HAVE UNDERGONE ENDOVASCULAR PROCEDURES UTILIZING UP TO 12F PROCEDURAL SHEATHS

ReliaSeal Protocol Number: P22-8301 Version: 3.0 Version Date: 31Jan2023

#### **Investigator Protocol Signature Page**

I have read this protocol and agree that it contains all necessary details for carrying out this study. I will conduct the study in accordance with the design and specific provisions outlined herein.

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure they are fully informed regarding the investigational product and the conduct of the study.

I will use the informed consent form approved by Sponsor and the IRB and will fulfill all responsibilities for submitting pertinent information to the IRB responsible for this study.

I also agree to report all information or data in accordance with the protocol and I agree to report any serious adverse events (SAE), and unanticipated adverse device effect (UADE) as defined in the protocol.

I further agree that Sponsor and/or designee have access to any original source documents from which case report form (CRF) information may have been generated.

I also agree to have control over all clinical supplies (including investigational product) provided by Sponsor and/or designees and collect and handle all clinical specimens in accordance with the protocol.

The below signed confirm herewith to have read and understood this study protocol and/or amendment and appendices; furthermore, to accomplish this study in accordance with the protocol, ICH/GCP guidelines, applicable international standards and all applicable country, local and federal regulations; and to accept respective revisions conducted by authorized personnel of Sponsor and by regulatory authorities.

| Principal Investigator | (print) | |
|------------------------|-------------|----------|
| Principal Investigator | (signature) | <br>Date |
| Institution Name/Locat | ion | |

100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




## **Table of Contents**

| Appro | oval Signatures | 2 |
|---|---|---|
| Invest | tigator Protocol Signature Page | 3 |
| Table | of Contents | 4 |
| Proto | col Synopsis | 8 |
| 1 | Study Management Team | 14 |
| 2 | Introduction | 15 |
| 2.1 | Product characteristics | 15 |
| 2.2 | Structural composition, operation principle and mechanism of action | 16 |
| 3 | Study Objectives | 16 |
| 4 | Indication | 17 |
| 5 | Contraindications | 17 |
| 6 | Precautions | 17 |
| 7 | Warnings | 17 |
| 8 | Benefits/Risks | 18 |
| 8.1 | Benefits | 18 |
| 8.2 | Risks | 18 |
| 9 | Study Design | 19 |
| 9.1 | Overview | 19 |
| 9.2 | Duplex Ultrasound sub-study | 19 |
| 10 | Study Population/Selection Criteria | 20 |
| 10.1 | Inclusion Criteria | 20 |
| 10.2 | Exclusion Criteria | 20 |
| | 10.2.1 Pre-procedural Exclusion Criteria | 20 |
| | 10.2.2 Intra-Procedural Exclusion Criteria | 21 |
| 11 | Study Endpoints | 22 |



100606833 | Rev:4 Released: 19 May 2023

## ReliaSeal / P22-8301

| 11.1 | Primary Endpoints | 22 |
|------|-----------------------------------------------------------------|----|
| | 11.1.1 Primary Safety Endpoint | 22 |
| | 11.1.2 Primary Effectiveness Endpoint | 22 |
| 11.2 | Secondary Endpoints | 22 |
| | 11.2.1 Secondary Safety Endpoint | 22 |
| | 11.2.2 Secondary Effectiveness Endpoints include the following: | 23 |
| 11.3 | Other/Additional Endpoints | 23 |
| 12 | Informed Consent | 23 |
| 13 | Screening and Enrollment | 25 |
| 13.1 | Screening Period | 25 |
| | 13.1.1 Screening Assessments | 25 |
| | 13.1.2 Screen Failures and Pre-screen Failures | 25 |
| 13.2 | Enrollment | 26 |
| 14 | Treatment Plan | 26 |
| 14.1 | Index Procedure | 26 |
| 14.2 | Post-Procedure Care/Discharge | 27 |
| 14.3 | Recommended Medication Regimen | 28 |
| 14.4 | Follow-up Visits/Assessments | 28 |
| 14.5 | Lost to Follow-up | 29 |
| 14.6 | Unscheduled Visits | 29 |
| 14.7 | Subject Early Discontinuation | 30 |
| 14.8 | Subject Study Completion | 30 |
| 15 | Adverse Event Reporting | 30 |
| 15.1 | Adverse Event | 30 |
| 15.2 | Serious Adverse Events | 31 |
| 15.3 | Unanticipated Adverse Device Effects | 32 |
| 15.4 | Sponsor Progress Reports | 32 |
| 16 | Statistics/Data Analyses | 32 |
| 16.1 | Randomization | 32 |



100606833 | Rev:4 Released: 19 May 2023

## ReliaSeal / P22-8301

| 16.2 | Device F | ailures and Malfunctions | 33 |
|---|---|---|---|
| 16.3 | Analysis Population | | |
| 16.4 | Statistical Hypotheses for Endpoints | | |
| 16.5 | Primary \$ | Safety Endpoint | 34 |
| 16.6 | Seconda | ry Safety Endpoint | 35 |
| 16.7 | Seconda | ry Effectiveness Endpoints | 36 |
| 16.8 | Sample 9 | Size Determination | 36 |
| 16.9 | Statistica | l Analysis Methods | 38 |
| | 16.9.1 | Primary Analysis | 39 |
| | 16.9.2 | Secondary Safety Analysis | 40 |
| | 16.9.3 | Secondary Efficacy Analyses | 40 |
| | 16.9.4 | Additional analysis | 41 |
| | 16.9.5 | Analysis of Roll-in Subjects | 41 |
| | 16.9.6 | Study site poolability | 41 |
| | 16.9.7 | Interim Analysis | 41 |
| 16.10 | )Sub-Gro | up Analysis | 42 |
| 16.11 | 1 Missing [ | Oata | 43 |
| 16.12 | 2Reportino | J | 43 |
| 17 | Quality | Control and Quality Assurance | 43 |
| 17.1 | Regulato | ry and Ethical Compliance | 43 |
| 17.2 | Data Qua | ality Assurance | 44 |
| 17.3 | Clinical E | Oata | 44 |
| 17.4 | Monitorin | ng | 45 |
| 17.5 | Protocol | Modifications | 46 |
| | 17.5.1 | Protocol Amendments | 46 |
| | 17.5.2 | Protocol Deviations/Noncompliance | 46 |
| | 17.5.3 | Emergency Deviations | 46 |
| 17.6 | Audits | | 46 |
| 17.7 | 7 Subject Confidentiality47 | | |
| 17.8 | 8 Institutional Review Board (IRB)47 | | |



100606833 | Rev:4 Released: 19 May 2023

### ReliaSeal / P22-8301

| 18 | Record Keeping/Publication Policy | 48 |
|-------|----------------------------------------------------|----|
| 18.1 | Record Retention | 48 |
| 18.2 | Use of Information and Publications | 48 |
| 19 | Investigational Product Accountability | 49 |
| 19.1 | Study Investigational Product Accountability | 49 |
| 19.2 | Instructions for Return of Investigational Product | 50 |
| 20 | Committees | 50 |
| 20.1 | Clinical Events Committee | 50 |
| 20.2 | Data and Safety Monitoring Board | 50 |
| 21 | Early Termination or Suspension | 51 |
| Appen | ndix A. Definitions | 53 |
| Appen | ndix B. Acronyms and Abbreviation | 55 |
| Appen | ndix C. References | 58 |

**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


A MULTICENTER, PROSPECTIVE, RANDOMIZED, CONTROLLED, OPEN LABEL TRIAL TO EVALUATE THE SAFETY AND EFFICACY OF MYNX CONTROL™ VENOUS VASCULAR CLOSURE DEVICE 6F12F VS. MANUAL COMPRESSION IN PATIENTS WHO HAVE UNDERGONE ENDOVASCULAR
PROCEDURES UTILIZING UP TO 12F PROCEDURAL SHEATHS

ReliaSeal Protocol Number: P22-8301 Version: 3.0 Version Date: 31Jan2023

## **Protocol Synopsis**

| femoral venous access sites in patients who have undergone endovascular procedures utilizing up to 12F, with single or multiple access sites in one or both limbs. Device Name MYNX CONTROL™ Venous Vascular Closure Device 6F-12F Device Model Number MX61260CL Device Category Class III medical device Current indication: MYNX CONTROL™ Vascular Closure Device is indicated for use to seal femoral arterial access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F, or 7F procedural sheath. Proposed expanded indication sought: The MYNX CONTROL™ Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural sheaths, with single or multiple access sites in one or both limbs. | Primary Objective | To demonstrate safety and efficacy of the MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression in sealing |
|---|---|---|
| access sites in one or both limbs. Device Name MYNX CONTROL™ Venous Vascular Closure Device 6F-12F Device Model Number Device Gategory Class III medical device Current indication: MYNX CONTROL™ Vascular Closure Device is indicated for use to seal femoral arterial access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F, or 7F procedural sheath. Proposed expanded indication sought: The MYNX CONTROL™ Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural sheaths, with single or multiple access sites in one or both limbs. Hypothesis Time to ambulation will be significantly less for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device than those using manual compression. Time to hemostasis will be at least 5 minutes less for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device than those using manual compression. Rate of combined major venous access site closure-related complications through 30 days post procedure for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. Study Design A multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. Study Design A multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device of F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. | | |
| Device Name MYNX CONTROL™ Venous Vascular Closure Device 6F-12F Device Model Number MX61260CL Device Category Class III medical device Indication for Use Current indication: | | |
| Device Model Number Device Category Class III medical device | | |
| Class III medical device | Device Name | MYNX CONTROL™ Venous Vascular Closure Device 6F-12F |
| Current indication: MYNX CONTROL™ Vascular Closure Device is indicated for use to seal femoral arterial access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F, or 7F procedural sheath. Proposed expanded indication sought: The MYNX CONTROL™ Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural sheaths, with single or multiple access sites in one or both limbs. Hypothesis | | |
| MYNX CONTROL™ Vascular Closure Device is indicated for use to seal femoral arterial access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F, or 7F procedural sheath. Proposed expanded indication sought: The MYNX CONTROL™ Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural sheaths, with single or multiple access sites in one or both limbs. Hypothesis Time to ambulation will be significantly less for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device than those using manual compression. Time to hemostasis will be at least 5 minutes less for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device than those using manual compression. Rate of combined major venous access site closure-related complications through 30 days post procedure for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. Study Design A multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. Number of Patients 204 patients (2:1 randomized - 136 VCD:68 manual compression) | | Class III medical device |
| The MYNX CONTROL™ Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural sheaths, with single or multiple access sites in one or both limbs. Hypothesis Time to ambulation will be significantly less for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device than those using manual compression. Time to hemostasis will be at least 5 minutes less for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device than those using manual compression. Rate of combined major venous access site closure-related complications through 30 days post procedure for patients treated with the MYNX CONTROL™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. Study Design A multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. Number of Patients 204 patients (2:1 randomized - 136 VCD:68 manual compression) | Indication for Use | MYNX CONTROL™ Vascular Closure Device is indicated for use to seal femoral arterial access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F, or 7F |
| MYNX CONTROL ™ Venous Vascular Closure Device than those using manual compression. Time to hemostasis will be at least 5 minutes less for patients treated with the MYNX CONTROL ™ Venous Vascular Closure Device than those using manual compression. Rate of combined major venous access site closure-related complications through 30 days post procedure for patients treated with the MYNX CONTROL ™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. Study Design A multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. Number of Patients 204 patients (2:1 randomized - 136 VCD:68 manual compression) | | The MYNX CONTROL™ Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural |
| with the MYNX CONTROL ™ Venous Vascular Closure Device than those using manual compression. Rate of combined major venous access site closure-related complications through 30 days post procedure for patients treated with the MYNX CONTROL ™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. Study Design A multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. Number of Patients 204 patients (2:1 randomized - 136 VCD:68 manual compression) | Hypothesis | |
| complications through 30 days post procedure for patients treated with the MYNX CONTROL ™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. Study Design A multicenter, prospective, randomized, controlled, open label clinical trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. Number of Patients complications through 30 days post procedure periodices with the MYNX Closure Device will be non-inferior to the rate for patients using manual compression. | | with the MYNX CONTROL ™ Venous Vascular Closure Device than |
| trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. Number of Patients 204 patients (2:1 randomized - 136 VCD:68 manual compression) | | complications through 30 days post procedure for patients treated with the MYNX CONTROL ™ Venous Vascular Closure Device will be non-inferior to the rate for patients using manual compression. |
| | Study Design | trial designed to evaluate safety and efficacy of use of MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression to seal femoral access sites in patients who have undergone endovascular procedures utilizing up to 12F procedural sheaths in one or both limbs. |
| Reference/Control Treatment Manual Compression | Number of Patients | 204 patients (2:1 randomized - 136 VCD:68 manual compression) |
| | Reference/Control Treatment | Manual Compression |

**Cordis** 

100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301


| Study Purpose | To demonstrate safety and efficacy of the MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression in sealing femoral venous access sites in patients who have undergone endovascular procedures utilizing one or more procedural sheaths up to 12F with single or multiple access sites in one or both limbs. |
|---|---|
| Study Centers | Approximately 15 study sites will participate in United States, with a minimum of 5 sites enrolling in the trial. |
| Duplex Ultrasound sub study | At select sites, a subset of 72 subjects (48 from the device group and 24 from the control group) will have an ultrasound examination of the access sites performed during the index procedure, at the time of discharge and at the 30 day (± 7 days) office visit (only for those subjects that have documented evidence of complications at the discharge ultrasound). |
| Eligibility Criteria | Inclusion Criteria: |
| | ALL patients must meet the following criteria prior to enrollment: |
| | <ol> <li>Age ≥18</li> <li>Able and willing to provide informed consent and to complete a follow-up visit at 30 ± 7 days</li> <li>Planned catheter-based procedures via the common femoral vein(s) using up 6F to 12F introducer sheaths which meet indications for elective, nonemergent interventions of disease state, without contraindications for emergent vascular surgery or manual compression of the venous access sites</li> </ol> |
| | Exclusion Criteria: |
| | Patients will be excluded if ANY of the following exclusion criteria apply: |
| | <ol> <li>Any use of systemic steroids (IV or oral) within 30 days of procedure</li> <li>History of deep vein thrombosis, pulmonary embolism, or thrombophlebitis within 6 months of procedure</li> <li>Presence of thrombocytopenia (platelet count &lt; 100,000 cells/mm3) or anemia (hemoglobin &lt; 10 g/dL, hematocrit &lt; 30%)</li> <li>History of bleeding disorders such as hemophilia or von Willebrand's disease</li> <li>Currently involved in any other investigational clinical trial</li> </ol> |
| | <ol> <li>Currently involved in any other investigational clinical than Documented history of uncontrolled hypertension (i.e., systolic blood pressure &gt; 180 mm Hg), or critical illness requiring intravenous vasopressors for blood pressure stabilization</li> <li>Femoral arteriotomy or venotomy in either limb within 10 days pre procedure</li> <li>Use of VCD in either limb within 30 days of procedure</li> <li>Any planned procedure involving femoral arterial or venous access in either limb within 30 days of procedure or prior to study exit</li> <li>Renal insufficiency (i.e., serum creatinine &gt; 2.5 mg/dL)</li> <li>Patients who are pregnant, planning to become pregnant during the study period, or lactating</li> <li>Body-mass index (BMI) &gt; 45 kg/m2 or &lt;20 kg/m2</li> </ol> |
| | 13.) Unable to routinely walk at least 20 feet without assistance |


**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


Known allergy/adverse reaction to polyethylene glycol or contrast medium 15.) Planned procedures (including staged) or concomitant conditions/comorbidities that per investigator's judgment may extend ambulation attempts beyond 2-3 hours, and/or require extended hospitalization or re-hospitalization 16.) Previous vascular surgery or repair in the vicinity of the target access site within the previous 90 days of the procedure 17.) Active systemic infection, or cutaneous infection or inflammation in the vicinity of the target access site 18.) Current COVID-19 infection (with or without symptoms), positive test for COVID- 19 within 14 days, or recent exposure to a person with COVID-19 infection 19.) Patients who refuse blood transfusion if it were to be needed 20.) Patients with expected life of less than 30 days Patients who meet ANY of the following criteria during the index procedure will be excluded: 1.) Any attempt at femoral arterial access or inadvertent arterial puncture with hematoma during the procedure 2.) Any procedural complications that may interfere with routine recovery, ambulation, or discharge eligibility times 3.) Physician deems that a different hemostasis approach for venous access sites is necessary Physician deems that the subject should not attempt protocol-4.) required ambulation (reference ambulation protocol per section 14.2) 5.) Venous access site location is noted to be above the inquinal ligament (cephalad to lower half of the femoral head or the inferior epigastric vein origin from the external iliac vein) 6.) Intra-procedural bleeding around sheath, or suspected intraluminal thrombus, hematoma, pseudoaneurysm, or AV fistula 7.) Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, accidental arterial stick with hematoma, "back wall stick", etc.) 8.) A < 6F or > 12F procedural sheath is present at any time during the procedure or at closure Primary Effectiveness Endpoint Primary Endpoint(s) Time to Ambulation (TTA): Defined as time (in hours) between removal of the MYNX CONTROL™ Venous Vascular Closure Device 6F-12F device (device group) or of the final sheath (control group) and when subject stands and walks 20 feet without evidence of rebleeding from any femoral venous access site. Time to Hemostasis (TTH): Defined as time (in minutes) between removal of each MYNX CONTROL™ Venous Vascular Closure Device 6F-12F device (device group) or of each sheath (control group) and first observed and confirmed venous hemostasis (per access site analysis)


**Cordis** 

100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301


| | Primary Safety Endpoint: |
|---|---|
| | Rate of CEC adjudicated combined <b>major</b> venous access site closure- related complications through 30 days post procedure, attributed directly to VCD or manual compression without other likely cause. • Access site-related bleeding requiring transfusion, surgical intervention, or rehospitalization • Vascular injury requiring surgical repair • Access site-related infection confirmed by culture and sensitivity, requiring intravenous antibiotics and/or extended hospitalization • New onset, permanent (i.e., persisting at 30-day follow-up) access site-related nerve injury • New onset access site-related nerve injury requiring surgical repair • Pulmonary embolism requiring surgical or endovascular intervention and/or resulting in death, to be confirmed by CT pulmonary angiography, lung ventilation/perfusion scan (VQ scan), or autopsy • Pulmonary embolism not requiring surgical or endovascular intervention and/or not resulting in death, to be confirmed by CT pulmonary angiography or lung ventilation/perfusion scan (VQ scan) |
| Secondary Endneint(s) | Secondary Safety Endpoint: |
| Secondary Endpoint(s) | Rate of CEC adjudicated combined minor venous access site closure related complications within 30 days post-procedure, attributed directly to VCD or manual compression without other likely cause. • Pseudoaneurysm – Treated with thrombin injection, fibrin adhesive injection, or ultrasound guided compression and documented by ultrasound • Pseudoaneurysm – Not requiring treatment • AV Fistula requiring treatment, documented by ultrasound • Av Fistula not requiring treatment, documented by ultrasound • Access site related hematoma > 6 cm documented by ultrasound • Access site-related bleeding requiring > 30 min to achieve hemostasis • Late access site-related bleeding (following hospital discharge eligibility) • Transient loss of ipsilateral lower extremity pulse • Ipsilateral deep vein thrombosis documented by ultrasound • Transient access site-related nerve injury • Access site vound dehiscence • Local access site infection confirmed by culture and sensitivity, treated with intramuscular or oral antibiotics – minor • Local access site inflammatory reaction – Minor • Allergic reaction • Ecchymosis |


Cordis

100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301

| | Secondary Effectiveness Endpoints: |
|---|---|
| | Time to Discharge Eligibility- defined as elapsed time (in hours) between removal of the final MYNX CONTROL™ Venous VCD (device group) or removal of the final sheath (control group) and when subject is eligible for discharge from the institution based on the assessment of the attending physician. |
| | Procedural Success: attainment of final hemostasis at all venous access sites without major venous access site closure-related complications through 30 days |
| | <ul> <li>Device Success (for device group): ability to successfully<br/>deploy the MYNX CONTROL™ Venous VCD delivery<br/>system, deliver the polyethylene glycol hydrogel sealant, and<br/>achieve hemostasis (device group only)</li> </ul> |
| Additional Endpoints | Pain score at time of discharge eligibility. |
| Sample Size | Total enrollment of 204 patients (2:1 randomized – 136 VCD: 68 manual compressions) |
| Duration of Subject<br>Participation | ALL patients will be followed through 30 days post procedure. Once all enrolled patients have completed follow-up, the study will be considered complete. |
| Statistics/Testing Methods | Data analysis will follow the intention-to-treat principle and will be conducted at the per access site or per patient level as indicated below, with a non-inferiority analysis for primary safety endpoint and superiority analyses for primary and powered secondary effectiveness endpoint. |



100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301

Table 1. Time and Event Schedule (Please refer to Section 14 for details)

| | Screening<br>(-30 to day<br>0) | At time of<br>Index<br>Procedure<br>(day 0) | Post-<br>Procedure/ | Pre-<br>discharge | 1-Month<br>(30 ± 7 days) |
|---|---|---|---|---|---|
| Informed consent (within 60 days of index procedure) | Х | | | | |
| Pre-op Inclusion / Exclusion Criteria Assessment | Х | | | | |
| Demographics | x | | | | |
| Physical exam/Medical History | Х | | | | Х |
| Laboratory Tests (PLT, WBC, HGB, HCT, creatinine, PT or INR) | X¹ | | | | Х |
| Intra-procedural Exclusion Criteria<br>Assessment | | X* | | | |
| Randomization | | Х | | | |
| Study Endpoint Data Collection: | | | | | |
| TTH determination | | Х | | | |
| TTA determination | | | X | | |
| TTDE determination | | | Х | | |
| Device Success | | Х | | | |
| Procedure Success | | | | | Х |
| Concomitant Medications (e.g., antiplatelet, anti-coagulant, anti-thrombotic agents, etc.) | х | Х | Х | | Х |
| Post Op Pain assessment | | | X | | |
| Adverse Events | | Х | Х | | Х |
| Ultrasound Exam (DUS substudy only) | | | | X ** | X *** |

<sup>&</sup>lt;sup>1</sup> Laboratory tests should be done within -7 to 0 days of index procedure

<sup>\*</sup> Intra-op inclusion/exclusion criteria will be evaluated once operator is able to visualize and assess sheath placement and the anatomy of all venous access sites
\*\* Ultrasound is required for subjects in the DUS sub-study only

<sup>\*\*\*</sup> Ultrasound may be required at 30 days if complication is observed on discharge DUS for subjects in DUS substudy



100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301


## 1 Study Management Team

## **Table 2: Study Management Team**

| Sponsor | Cordis US Corp |
|---------------------------------|---------------------|
| Medical Monitor | Nusrath Sultana, MD |
| National Principal Investigator | Javier Sanchez, MD |
| Monitoring | NAMSA |
| Data Management | Medrio |
| Safety Management | NAMSA |
| Statistics | NAMSA |
| Medical Writing | NAMSA |
| Duplex Ultrasound Core Lab | NAMSA |

Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


#### 2 Introduction

Techniques for closure of an arteriotomy or venotomy site have evolved from direct suture-based surgical closure to the use of VCDs. VCDs were developed in the 1990s with the aim of achieving hemostasis efficiently in a way that is satisfactory to the patient with limited complications.<sup>9, 10</sup> Ideally, VCDs should safely attain complete hemostasis, close the access site regardless of the size, and this should be achievable even with the use of anticoagulants.<sup>9</sup>

The target patient population indicated for VCDs are patients undergoing diagnostic and/or interventional procedures involving access to the coronary or peripheral vascular system and patients with contraindications to undergo surgery due to operative risk and comorbidities. Following percutaneous vascular access, VCDs are used to achieve hemostasis after interventional or diagnostic endovascular procedures. VCDs, such as the MYNX VCD Product Family and EXOSEAL VCD Product Family provide a method of achieving hemostasis at the femoral access sites in patients who have undergone endovascular procedures utilizing a 5F, 6F, or 7F procedural sheath. These procedures are generally performed by physicians from a broad range of medical specialties to include interventional radiology, vascular surgery, and cardiology, as well as smaller subspecialists trained in the application of endovascular techniques. For this study, we have expanded the indication of the MYNX CONTROL VCD to include up to 12F procedural sheath for femoral venous access. Procedures treated using this larger bore sheath include, but are not limited to, cardiac ablations, structural heart procedures, and cardiac interventions.

The traditional and most used alternative to VCDs is manual compression (MC). MC is considered the standard of care and is relied upon either primarily or when VCDs fail. MC is labor-intensive and results in considerable discomfort for the patient. Meta-analyses comparing MC to VCDs showed that with MC there was an increase in time-to-hemostasis (TTH), time-to-ambulation (TTA). <sup>15, 16</sup> An increased risk of hematoma formation was associated with MC. <sup>15</sup> The rate of complications was comparable between VCDs and MC (12% for VCDs and 13% for MC), however, major complications were lower in the VCD group. <sup>16</sup> VCDs were associated with a low risk of infection and thrombosis (0.6% for infection; 0.3% for thrombosis). <sup>16</sup>

The MYNX CONTROL™ Venous Vascular Closure Device (VCD) is indicated for use to seal femoral arterial access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing a 5F, 6F or 7F procedural sheath.

#### 2.1 Product characteristics

The MYNX CONTROL™ Venous Vascular Closure Device (VCD) is designed to achieve femoral vein hemostasis via delivery of the GRIP TECHNOLOGY™ sealant, an extravascular, water-soluble synthetic hydrogel, using a balloon catheter in conjunction with a standard procedural sheath. The GRIP TECHNOLOGY™ sealant is made of a polyethylene glycol (PEG) material which expands upon contact with blood and subcutaneous fluids. Refer to Figure 1 (below).


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


#### 2.2 Structural composition, operation principle and mechanism of action

The MYNX VCD product family are designed to achieve hemostasis of femoral access sites following diagnostic or interventional endovascular procedures. Hemostasis is accomplished via delivery of an extravascular polyethylene glycol (PEG) sealant using a balloon catheter (delivery system) in conjunction with a standard procedural sheath. Upon contact with blood and subcutaneous fluids, the sealant expands and adheres to the arteriotomy or venotomy to achieve hemostasis. The sealant is resorbed by the body within 30 days.

The design of the MYNX CONTROL™ Venous VCD is based on the design of the current MYNX CONTROL™ VCD (arterial). The only difference in design is the Sheath Catch. The Sheath Catch facilitates the withdrawal of the 6F/7F Catheter Sheath Introducer (CSI) from the tissue tract during the withdrawal of the MYNX CONTROL™ VCD (current). This is achieved by a distal hook which latches onto the sideport on the CSI. The proposed sheath catch design on the MYNX CONTROL™ Venous VCD will be based on the current design but will allow larger CSIs (up to 12F) to fit into the Sheath Catch. Like the current Sheath Catch design, connection to the CSI will be achieved with a distal hook and be universally compatible with the leading CSI brands on the market.



Figure 1: MYNX CONTROL™ Venous Vascular Closure Device 6F-12F

## 3 Study Objectives

To demonstrate safety and efficacy of the MYNX CONTROL™ Venous Vascular Closure Device 6F-12F vs. manual compression in sealing femoral venous access sites in patients who have undergone endovascular procedures utilizing one or more procedural sheaths up to 12F.


100606833 | Rev:4 Released: 19 May 2023




#### 4 Indication

ReliaSeal / P22-8301

Proposed Indications for Use:

The MYNX CONTROL™ Venous VCD 6F-12F is indicated for use to seal femoral venous access sites while reducing times to hemostasis and ambulation in patients who have undergone diagnostic or interventional endovascular procedures utilizing 6F to 12F procedural sheaths, with single or multiple access sites in one or both limbs.

#### 5 Contraindications

There are no known contraindications for the MYNX CONTROL™ Venous Vascular Closure Device 6F-12F.

#### 6 Precautions

The MYNX CONTROL™ Venous VCD should only be used by a trained licensed physician or healthcare professional. The MYNX CONTROL™ Venous VCD should not be used in patients with a known allergy to PEG. The MYNX CONTROL™ Venous VCD should not be used with sheaths longer than 12 cm effective length or incompatible sheaths listed in **Table 3.** Exposure to temperatures above 25°C (77°F) may damage the components.

Table 3

| MANUFACTURER | DESCRIPTION |
|--------------|----------------------------------|
| Cook | Check-Flo® Performer® Introducer |

## 7 Warnings

Do not use if components or packaging appear to be damaged or defective or if any portion of the packaging has been previously opened. DO NOT REUSE OR RESTERILIZE. The MYNX CONTROL™ Venous VCD 6F-12F is for single use only. The catheter is loaded with a single Hydrogel sealant. Reuse of the device would result in no delivery of Hydrogel sealant. Reuse of this product, including after reprocessing and/or re-sterilization, may cause a loss of structural integrity which could lead to a failure of the device to perform as intended and may lead to a loss of critical labeling/use information all of which present a potential risk to patient safety. Do not use the MYNX CONTROL™ Venous VCD 6F-12F if the puncture site is located above the inguinal ligament based upon bony landmarks, since such a puncture site may result in a hematoma/bleed. Perform a femoral venogram (as applicable) to verify the location of the puncture site. Do not use the MYNX CONTROL™ Venous VCD 6F-12F if the puncture is through the posterior wall as such punctures may result in a retroperitoneal hematoma/bleed.



100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


#### 8 Benefits/Risks

#### 8.1 Benefits

There are several resource and time saving benefits associated with the use of VCDs. Time-to-hemostasis (TTH), time-to-ambulation (TTA) and time-to-discharge eligibility(TTDE) have all been reported to be reduced with the use of VCDs. To Meta-analyses of RCTs showed that that TTH was significantly shorter with VCDs compared to MC. The total number of NC. The sequence of RCTs showed that that TTH was significantly reduced by using VCDs compared to MC. The total number of NC. The number of NC. The total number of NC. The number of NC. T

As per clinical study data available for CORDIS VCDs, the devices provide an acceptable risk/benefit profile. Based on the clinical study data accumulated to evaluate the safety and effectiveness of these devices, the results for clinical studies show excellent rates of technical success and reduced time to hemostasis, ambulation, and discharge for the CORDIS VCDs. This indicates that with the use of these devices, patients have the potential to experience significant clinical improvements.

The potential benefits of the MYNX CONTROL™ Venous VCD for 6-12F over manual compression alone to achieve venous hemostasis have not yet been proven and outcomes will be evaluated because of this trial.

#### 8.2 Risks

The most serious recognized risks associated with femoral vessel closure procedures occur rarely and include, but are not limited to, the following:

- Vascular injury requiring repair
- New onset, permanent (i.e., persisting at 30-day follow-up) access site-related nerve injury
- Bleeding or hematoma at any venous access site requiring transfusion, surgical intervention, or re-hospitalization
- New ipsilateral lower extremity ischemia requiring invasive/non-invasive intervention
- Generalized access site related infection requiring intravenous antibiotics and/or extended hospitalization
- Retroperitoneal bleed


ReliaSeal / P22-8301




- Vessel Occlusion
- Pulmonary embolism
- Death

Other less serious potential risks (can be managed clinically or pharmaceutically) are included, but are not limited to, the following:

- Pseudoaneurysm Treated with thrombin injection
- Pseudoaneurysm Not requiring treatment
- AV Fistula
- Hematoma > 6 cm
- Access site-related bleeding requiring > 30 min to achieve hemostasis
- Late access site-related bleeding (following hospital discharge)
- Ipsilateral lower extremity arterial emboli
- Transient loss of ipsilateral lower extremity pulse
- Ipsilateral deep vein thrombosis
- Transient access site-related nerve injury
- Access site-related vessel laceration
- Local access site infection Minor
- Local access site inflammatory reaction Minor
- Allergic reaction
- Ecchymosis

### 9 Study Design

#### 9.1 Overview

This study is a multicenter, prospective, randomized, controlled, open label clinical study to enroll 204 patients with an additional group of patients to be part of the initial roll-in phase. The 204 patients will be randomized to either a device arm or a manual compression arm using a 2:1 randomization scheme (136 MYNX CONTROL™ patients and 68 manual compression patients). Two (2) roll-in patients per physician will be allowed. All patients who sign the informed consent and randomized to either treatment group will be followed through 30 days post procedure. There will be up to 15 participating study sites, with a minimum of five (5) sites, all located in the United States. Details of the randomization and roll-in process can be found in section 16.1. Each study site will be limited to enrolling a maximum of 45 subjects.

#### 9.2 Duplex Ultrasound sub-study

A sub-study of this pivotal U.S. clinical trial will be performed utilizing independent analysis of non-invasive duplex ultrasound (DUS) imaging in 48 device subjects and 24 MC subjects predischarge and potentially again at the 30-day follow-up if an observation of a complication occurred on the pre-discharge ultrasound. Specific investigational sites will be designated as ultrasound sites. These sites will include subjects in the ultrasound subset imaging until a total of 72 patients have been evaluated in both groups. Informed consent will be obtained from all


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


subjects participating in this sub-study. All sub-study sites will be instructed to perform duplex ultrasonography of the femoral vascular structures. Images will be uploaded and interpreted by an independent core lab. NAMSA is the core lab for this sub study.

NAMSA 4 World Trade Center 150 Greenwich Street, 49<sup>th</sup> FL New York, NY 10007

#### 10 Study Population/Selection Criteria

The following outline the specific inclusion and exclusion criteria for the study. Before the study randomization, a patient must meet all the inclusion and no exclusion criteria.

Prior to any study-specific activities, all patients must sign and date the most current IRB-approved Informed Consent Form (ICF).

#### 10.1 Inclusion Criteria

Patients must meet ALL the following inclusion criteria to be enrolled in the study:

- 1. Age >18
- 2. Able and willing to provide informed consent and to complete a follow-up visit at 30 days
- Planned catheter-based procedures via the common femoral vein(s) using up 6F to 12F introducer sheaths which meet indications for elective, nonemergent interventions of disease state, without contraindications for emergent vascular surgery or manual compression of the venous access sites

#### 10.2 Exclusion Criteria

Patients will be excluded if they meet ANY of the following exclusion criteria:

#### 10.2.1 Pre-procedural Exclusion Criteria

Patients who meet any of the following criteria before the index procedure will be excluded:

- 1. Any use of systemic steroids (IV or oral) within 30 days of procedure
- History of deep vein thrombosis, pulmonary embolism, or thrombophlebitis within 6 months of procedure
- 3. Presence of thrombocytopenia (platelet count < 100,000 cells/mm3) or anemia (hemoglobin < 10 g/dL, hematocrit < 30%)
- 4. History of bleeding disorders such hemophilia or von Willebrand's disease
- 5. Currently involved in any other investigational clinical trial
- 6. Documented history of uncontrolled hypertension (i.e., systolic blood pressure > 180 mm Hg), or critical illness requiring intravenous vasopressors for blood pressure stabilization
- 7. Femoral arteriotomy or venotomy in either limb within 10 days pre procedure


100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




- 8. Use of VCD in either limb within 30 days of procedure
- 9. Any planned procedure involving femoral arterial or venous access in either limb within 30 days or prior to study exit
- 10. Renal insufficiency (i.e., serum creatinine > 2.5 mg/dL)
- 11. Patients who are pregnant, planning to become pregnant during the study period, or lactating
- 12. Body-mass index (BMI) > 45 kg/m2 or <20 kg/m2
- 13. Unable to routinely walk at least 20 feet without assistance
- 14. Known allergy/adverse reaction to polyethylene glycol or contrast medium
- 15. Planned procedures (including staged) or concomitant conditions/comorbidities that per investigator's judgment may extend ambulation attempts beyond 2-3 hours, and/or require extended hospitalization or re-hospitalization
- 16. Previous vascular surgery or repair in the vicinity of the target access site within the previous 90 days of the procedure
- 17. Active systemic infection, or cutaneous infection or inflammation in the vicinity of the target access site
- 18. Current COVID-19 infection (with or without symptoms), positive test for COVID-19 within 14 days, or recent exposure to a person with COVID-19 infection
- 19. Patients who refuse blood transfusion if it were to be needed
- 20. Patients with expected life of less than 30 days

#### 10.2.2 Intra-Procedural Exclusion Criteria

Patients who meet any of the following criteria during the index procedure will be excluded:

- 1. Any attempt at femoral arterial access or inadvertent arterial puncture with hematoma during the procedure
- 2. Any procedural complications that may interfere with routine recovery, ambulation, or discharge eligibility times
- 3. Physician deems that a different hemostasis approach for venous access sites is necessary
- 4. Physician deems that the subject should not attempt protocol required ambulation (reference ambulation protocol per section 14.2)
- 5. Venous access site location is noted to be above the inguinal ligament (cephalad to lower half of the femoral head or the inferior epigastric vein origin from the external iliac vein)
- 6. Intra-procedural bleeding around sheath, or suspected intraluminal thrombus, hematoma, pseudoaneurysm, or AV fistula
- 7. Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, accidental arterial stick with hematoma, "back wall stick", etc.)
- 8. A < 6F or > 12F procedural sheath is present at any time during the procedure or at closure




100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


## 11 Study Endpoints

- 11.1 Primary Endpoints
- 11.1.1 Primary Safety Endpoint

Rate of CEC adjudicated combined **major** venous access site closure-related complications through 30 days post procedure, attributed directly to VCD or manual compression without other likely cause.

- Access site-related bleeding requiring transfusion, surgical intervention, or rehospitalization
- Vascular injury requiring surgical repair
- Access site-related infection confirmed by culture and sensitivity, requiring intravenous antibiotics and/or extended hospitalization
- New onset, permanent (i.e., persisting at 30-day follow-up) access site-related nerve injury
- · New onset access site-related nerve injury requiring surgical repair
- Pulmonary embolism requiring surgical or endovascular intervention and/or resulting in death, to be confirmed by CT pulmonary angiography, lung ventilation/perfusion scan (VQ scan), or autopsy
- Pulmonary embolism not requiring surgical or endovascular intervention and/or not resulting in death, to be confirmed by CT pulmonary angiography or lung ventilation/perfusion scan (VQ scan)
  - 11.1.2 Primary Effectiveness Endpoint

<u>Time to Ambulation (TTA)</u>: Defined as elapsed time (in hours) between removal of the MYNX CONTROL™ Venous Vascular Closure Device 6F-12F device (device group) or of the final sheath (control group) and when subject stands and walks 20 feet without evidence of rebleeding from any femoral venous access site.

<u>Time to Hemostasis (TTH):</u> Defined as elapsed time (in minutes) between removal of each MYNX CONTROL™ Venous Vascular Closure Device 6F-12F device (device group) or of each sheath (control group) and first observed and confirmed venous hemostasis (per access site analysis).

- 11.2 Secondary Endpoints
- 11.2.1 Secondary Safety Endpoint

Rate of CEC adjudicated combined **minor** venous access site closure related complications within 30 days post-procedure, attributed directly to VCD or manual compression without other likely cause. Types of minor complications include:


100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




- Pseudoaneurysm Treated with thrombin injection, fibrin adhesive injection, or ultrasound guided compression and documented by ultrasound
- Pseudoaneurysm Not requiring treatment
- Arteriovenous fistula requiring treatment, documented by ultrasound
- Arteriovenous fistula not requiring treatment, documented by ultrasound
- Access site-related Hematoma > 6 cm documented by ultrasound
- Access site-related bleeding requiring > 30 min to achieve hemostasis
- Late access site-related bleeding (following hospital discharge eligibility)
- Transient loss of ipsilateral lower extremity pulse
- Ipsilateral deep vein thrombosis documented by ultrasound
- Transient access site-related nerve injury
- Access site-related vessel laceration
- Access site wound dehiscence
- Localized access site infection confirmed by culture and sensitivity, treated with intramuscular or oral antibiotics—Minor,
- Local access site inflammatory reaction Minor
- Allergic reaction
- Ecchymosis

#### 11.2.2 Secondary Effectiveness Endpoints include the following:

<u>Time to Discharge Eligibility:</u> defined as elapsed time (in hours) between removal of the final MYNX CONTROL™ Venous Vascular Closure Device 6F-12F device (device group) or removal of the final sheath (control group) and when subject is eligible for discharge from the institution based on the assessment of the attending physician.

<u>Procedural Success</u>: attainment of final hemostasis at all venous access sites without major venous access site closure-related complications through 30 days.

<u>Device Success (for device group)</u>: ability to successfully deploy the MYNX CONTROL™ Venous VCD delivery system, deliver the polyethylene glycol hydrogel sealant, and achieve hemostasis (device group only).

#### 11.3 Other/Additional Endpoints

 Venous access site related pain at time of discharge eligibility measured by pain scores

#### 12 Informed Consent

Written Informed Consent must be obtained for all patients who are potential study candidates. Patients who meet pre-op inclusion/exclusion entry criteria will be invited to participate, and asked to sign the study-specific, Institutional Review Board (IRB)-approved Informed Consent form


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


before any study-specific tests or procedures are performed which are not standard-of-care. The study team shall follow all steps below when obtaining Informed Consent:

- 1. Provide each prospective subject/legal representative with a full explanation of the study (including all potential benefits and risks) and the informed consent form (ICF).
  - a. The informed consent form (ICF) should enable the subject or legal representative to understand:
    - the nature, objectives, benefits, implications, risks, and inconveniences of the clinical investigation
    - the subject's rights and guarantees regarding his/her protection, his/her right to refuse to participate in and the right to withdraw from the clinical investigation at any time without any resulting detriment and without having to provide any justification
    - the conditions under which the clinical investigation is to be conducted, including the expected duration of the subject's participation in the clinical investigation; and the possible treatment alternatives, including the follow-up measures if the participation of the subject in the clinical investigation is discontinued.
  - b. The ICF shall:
    - Be comprehensive, concise, clear, relevant, and understandable to the subject or legal representative
    - Be provided in a prior interview with a member of the clinical investigation team who is appropriately qualified under national law and delegated to this responsibility; gives special attention to the information needs of specific patient populations and individual patients as well as to the methods used to provide the information; verifies the subject has understood the information
    - Include information about an applicable damage compensation system; and
    - Include the unique, study identification number and information about the availability of clinical study results to the subject, to the extent possible, via a clinical study report and summary presented in terms understandable to the intended user, irrespective of the outcome of the clinical study.
- 2. Allow the prospective subject/legal representative to read the most current IRB approved informed consent form (ICF) and address any/all their questions.
- Obtain written consent (signature and date on the ICF) from the prospective subject/legal representative after the Investigator and/or designee is assured they understand all implications of participating in the study.


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


A copy of the ICF signed by the subject/legal representative and the Investigator and/or designee obtaining consent will be provided to the subject. In addition to the most current, IRB-approved ICF, the subject/legal representative must provide a signed HIPAA authorization and any other locally required documents, as applicable.

The Investigator and/or designee must clearly document the process for obtaining informed consent, including the date/time of obtaining consent, in the subject's medical record. It is the Investigator's responsibility to ensure that the informed consent process is performed in accordance with ICH-GCP applicable international standards and all applicable local and federal regulations.

Documented informed consent must be obtained within 60 days prior to the index procedure.

Exceptions to obtaining documented informed consent prior to the initiation of study-specific procedures would be in cases where necessary to eliminate an immediate apparent hazard and protect the life or physical well-being of a study subject.

## 13 Screening and Enrollment

- 13.1 Screening Period
- 13.1.1 Screening Assessments

In addition to obtaining written consent, the following assessments must be performed, and the subject verified to meet all pre-procedural inclusion criteria and none of the exclusion criteria prior to the procedure.

- 1) **Demographic Data**: Including but not limited to age, sex, weight, height, and race.
- 2) **Medical/Surgical History**: (30 days prior to the procedure) Review and documentation of subject's medical history, allergy assessment and risk factors.
- Physical Examination: Assessment per sites Standard of Care and to include collection of concomitant med and Laboratory Evaluations as below, height, weight, and BMI
- 4) **Concomitant Medications:** Peri-procedural medications that are taken within 24 hours of the procedure that may affect bleeding (e.g., anti-platelet, anti-coagulant, anti-thrombotic agents, etc.) will be documented
- 5) **Laboratory Evaluations:** (within one week prior to index procedure):
  - blood routine examination (PLT, WBC, HCT, HGB, and creatinine),
  - coagulation function (prothrombin time (PT) or INR),
  - pregnancy testing for women with fertility.
- 13.1.2 Screen Failures and Pre-screen Failures

Any consented patient who is confirmed to <u>not</u> qualify for study participation according to the eligibility criteria will be considered a screen failure and will neither be treated with the


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


investigational device nor be followed per protocol. Signed informed consent forms and all applicable documentation including source records indicating rationale for screen failure classification and screening logs will be reviewed during monitoring visits for all screen failure patients.

Pre-screen failures are defined who are confirmed as patients to not qualify for study participation according to the eligibility criteria after review their medical records (i.e. prior to providing informed consent). Such patients will neither treated with the study devices nor followed per protocol.

#### 13.2 Enrollment

The subject will be enrolled into the study at the end of the index procedure and once all procedural sheaths are in place under imaging guidance. It is at this time that the anatomy of all venous access sites is evaluated, and intra-procedural eligibility criteria can be verified. Each venous access site must meet all intra-procedural access site-specific criteria for the subject to be eligible. Once it has been determined that the subject does not meet any of the general intra-operative exclusion criteria, and that none of the venous access sites meet the specific access site exclusion criteria, then the subject is eligible for randomization.

#### 14 Treatment Plan

#### 14.1 Index Procedure

The Instructions for Use (IFU) provides detailed information on the product, safety, storage, design, deliverability, and sizing specifications. All information within the IFU should be referenced prior to each procedure and implantation of the study device.

If a subject is randomized to receive manual compression, it should be performed according to the institution's standard of care practice. If protamine is administered, the Investigator should follow institutional practice guidelines for re-checking ACT levels and/or waiting a specified time or for a target ACT value prior to removal of sheaths and application of manual compression.

If a subject is on Warfarin, any pre-procedure standard of care requirements should be followed.

#### The following will be collected at the time of the procedure:

- A0: Time of first index procedure sheath insertion
- A1 Time: time of removal of final index procedure device
- Sheath sizes used during procedure
- For each access site, the following should be recorded:
  - Access site location (left/right leg and location with respect to 2<sup>nd</sup> access site, if applicable)
  - HX.1 Time: time of removal of MYNX CONTROL<sup>™</sup> Venous device (device group) or removal of sheath (control group)


100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




- HX.2 Time: time venous hemostasis is achieved.
- Confirm venous hemostasis is maintained at 5 min after recorded hemostasis time (HX.2)
- Use of adjunctive compression (e.g., light manual compression, sandbags, or mechanical compression devices)

#### 14.2 Post-Procedure Care/Discharge

Following the index procedure, the site will notify the Sponsor of the subject enrollment status within the study database

#### The following will be documented after the procedure:

- A2 Time: Date and time the subject was able to ambulate 20 feet without venous rebleeding from the access site(s).
- 2. **A3 Time:** Date and time the subject is eligible for discharge based on the assessment of the attending physician or delegate.
- 3. A4 Time: Date and time the subject was discharged.
- 4. Concomitant Medications: Peri-procedural medications that are taken within 24 hours of the procedure that may affect bleeding (e.g., anti-platelet, anti-coagulant, anti-thrombotic agents, etc.) will be documented
- 5. Adverse event monitoring, including labs as per standard of care to assess any adverse event
- 6. Time to Ambulation- Defined as time (in hours) between removal of the final VCD (device group) or of the final sheath (control group) and when subject stands and walks 20 feet without evidence of rebleeding from any femoral venous access site.

NOTE: Since TTA is a primary effectiveness endpoint, the following ambulation guidelines apply to both groups.

- For the device group, ambulation must be attempted within 2-2.5 hours from time of final VCD removal. The groin should be checked every 15 minutes to verify status. Any ambulation delay beyond 2.5 hours will be considered a protocol deviation unless it is medically justified and documented.
- For the control group, institutional guidelines should be followed for ambulation. The groin should be checked every 15 minutes to verify status. Reasons for any ambulation delays beyond the institution's standard of practice should be documented.
- 7. Time to Discharge Eligibility- defined as elapsed time between removal of the final MYNX CONTROL™ Venous VCD (device group) or removal


**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


of the final sheath (control arm) and when subject is eligible for discharge from the institution based on the assessment of the attending physician or delegate. (Per-patient analysis)

- 8. Pain scale assessment
- 9. Duplex Ultrasound (pre-discharge) for those patients enrolled in DUS sub-study

NOTE 1: If there is any sign of active bleeding at the access site(s) after ambulation, measures should be taken to re-achieve hemostasis and then the subject re-ambulated when the Investigator determines that it is appropriate to do so. In these cases, TTA and TTDE will be repeated and documented when successful, and the re-bleeding will be documented as an adverse event.

NOTE 2: TTDE is not intended to impact the actual discharge time of the subjects from the hospital. Any delay of this discharge eligibility determination (i.e. >30 minutes following successful ambulation) unrelated to access site(s) assessment will be documented as a protocol deviation.

#### 14.3 Recommended Medication Regimen

Discharge medication should be administered per institutions standard of care and at the discretion of the Investigator. Details of this regimen must be recorded in the appropriate Case Report Form.

#### 14.4 Follow-up Visits/Assessments

All subjects will be required to complete a 30±7-day follow-up. The follow-up will include the following assessments:

- 1) **Concomitant Medications:** Peri-procedural medications that are taken within 24 hours of the procedure that may affect bleeding (e.g., anti-platelet, anti-coagulant, anti-thrombotic agents, etc.) will be documented
- 2) Laboratory Evaluations:
  - blood routine examination (PLT, WBC, HCT, HGB and creatinine),
  - coagulation function (prothrombin time (PT) or INR)
- 3) Adverse event monitoring
- 4) Duplex Ultrasound: for those subjects included in the DUS sub-study where a documented access site complication has been observed on the Discharge Ultrasound. Subjects should have their ultrasound appointments scheduled to ensure compliance.

NOTE: Every effort should be made to complete the required 30-day follow-up assessments on-site. If the subject is unable to complete an on-site 30-day follow-up, visit may be conducted by phone. If visit is conducted via phone, concomitant medications and safety information should be collected from subject or from subject's friend/family, if possible. Regardless, if visit is on-site or via phone, every


100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




attempt should be made to acquire all study assessments (including lab evaluations).

For DUS subset study – this must be obtained on-site. If visit is out of window to obtain DUS, document this as protocol deviation.

A Protocol Deviation will need to be completed for all study subjects who do not complete all 30-day follow-up visit assessments. If the missed visit is COVID-related, it will be categorized as such in the protocol deviation.

#### 14.5 Lost to Follow-up

For all active subjects, the site must first make three (3) contact attempts to reach the subject. If unsuccessful, the Investigator must then send a certified letter to the subject. All contact attempts must be adequately documented in the subject's source documents. When possible, the subject's primary care physician should also be asked for assistance with contacting the subject.

The subject will be considered lost to-follow-up only under the following circumstances:

- The site learns that all methods of contacting the subject are no longer viable (e.g., telephone number not in service, no forwarding address provided, no current/correct contact information available from the subject's primary care physician).
- Failure to reach/hear from the subject for the final protocol-required follow-up visit after all required contact attempts have been made.

#### 14.6 Unscheduled Visits

Unscheduled follow-up visits may be required to evaluate a subject from time to time to ensure the safety of study subjects. All complications and adverse events will be evaluated by the Investigator and reported according to Sponsor and IRB regulations.

If an unscheduled follow-up visit is required, the site study team will assess if the subject has undergone any interventional treatment or experienced any adverse events since the last protocol specified visit and will record such information on the appropriate CRF pages. All relevant information required to assess the event should be maintained in the subject's medical records and all relevant documentation required for event adjudication should be provided as requested by the Sponsor.

The following assessments may need to be completed at an unscheduled visit:

- Concomitant medications
- Physical examination
- Duplex Ultrasound (for subjects in the DUS sub-study with complications at discharge DUS)
- Adverse event monitoring
- Laboratory evaluations (see follow-up visit assessments in section 14.4)


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


#### 14.7 Subject Early Discontinuation

Every subject should be encouraged to remain in the study until they have completed the final, protocol-required follow-up visit at 30 days +/- 7 days post-discharge. If subject participation is prematurely discontinued, the reason for such must be documented in the subject's source documents and the CRF. Possible reasons for a subject's early exit from the study may include, but are not limited to, the following:

- Withdrawal of consent Subject decides to withdraw from the study. This
  decision must be "independent" (i.e., made by the subject) and documented in
  the subject's source records and the CRF. The reason for withdrawal of consent
  should also be inquired from the subject and documented if provided.
- Physician discretion The Investigator may choose to withdraw a subject from the study for reasons which include, but are not limited to, safety concerns.
- Death
- Lost to follow-up all methods of contacting the subject are no longer viable or the subject is unable to be reached to complete the 30-day follow-up visit.

Subjects who discontinue from the study early will not be replaced. Subjects who withdraw voluntarily or are withdrawn from the study per Investigator discretion cannot re-enter the study. The investigator(s)/institution(s) should arrange for any continued safety monitoring, treatment and/or follow-up of subjects who withdraw/are withdrawn from the study or determined as lost to follow-up as per standard-of-care/best clinical judgement. The Investigator can use existing data and may ask for the subject's permission to collect follow-up data about status and/or condition, including information related to the device performance, effectiveness, or safety. If permission is granted, the relevant data will be included in the clinical study report.

#### 14.8 Subject Study Completion

The clinical study will be considered complete when the last enrolled subject has completed the 30-day follow-up visit or protocol-required assessment. The sponsor will provide end-of-study notification to all participating sites for submission to their IRBs.

#### 15 Adverse Event Reporting

Any person who identifies an event or information that could impact subjects', users', or other persons' safety has an obligation to inform the Investigator and the sponsor of their concerns.

#### 15.1 Adverse Event

An Adverse Event (AE) is any untoward medical occurrence in a subject, whether anticipated or unanticipated. All AEs are reported from the subject's start time of enrollment until their exit from the study (i.e., point of study completion or premature discontinuation). AEs will be recorded and followed until resolution or stabilization of the event or until the subject has exited the study.


Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


Anyone should be encouraged to report AEs immediately upon awareness and may volunteer information at any time. At each evaluation, the Investigator will assess if an adverse event has occurred and will obtain all information required to complete the appropriate AE CRF(s). If an event occurs at an outside institution, the Investigator should obtain all or as much of the required AE information as possible.

For each AE, the Investigator should report at a minimum, the term/description, start/end dates, severity, serious/non-serious classification, treatment, and outcome of the AE and determine its causality/association to the investigational product or procedures involved in the clinical study.

All sites will be trained on severity and causality of AEs and completing the AE Case Report Form

#### 15.2 Serious Adverse Events

A Serious Adverse Event (SAE) is a type of AE and defined as any untoward medical occurrence that:

- a) Led to a death
- b) Led to a serious deterioration in the health of the subject that
  - Results in a life-threatening illness or injury
  - Results in a permanent or significant impairment of a body structure or a body function
  - Requires hospitalization or prolongation of existing hospitalization
  - Results in an important medical event which jeopardizes the subject and may require medical or surgical intervention to prevent permanent impairment to a body structure or one of the above outcomes
- c) Led to fetal distress, fetal death or a congenital abnormality or birth defect

The Investigator must report all SAEs to the Sponsor and/or designee by any applicable method within 24 hours or one working day of first awareness of the event by the study team at the institution and provide any additional information as required by the Sponsor/designee. The Electronic Data Capture (EDC) system should be the principal system used in reporting these events, if possible. In the case of death, all available information, e.g., autopsy or other postmortem findings, including causality/association to the investigational product, should be provided. The medical monitor of this study will decide if more follow-up information is needed in case the event is not resolved at the time of subject exit from the study.

The Investigator shall notify their IRB of SAEs which occurred at their site in accordance with their institutional requirements.

SAEs will be recorded and followed until resolution or stabilization of the event or until the subject has exited the study.


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


In the case of death, all available information, e.g., autopsy or other post-mortem findings, including causality/association to the investigational product, should be provided.

#### 15.3 Unanticipated Adverse Device Effects

An unanticipated adverse device effect (UADE) is defined as any serious adverse effect on health or safety or any life-threatening problem or death caused by or associated with an investigational product, if that effect, problem or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with an investigational product that relates to the rights, safety, or welfare of patients.

Potential UADEs occurring during the study must be reported by the Investigator to the Sponsor [through the EDC system or by other available means within 24 hours or one working day of first awareness of the event by the study team at the institution.

- If the Sponsor confirms the reported event qualifies as a UADE and presents as an
  unreasonable risk(s) to study subjects, they will terminate the entire study, or parts of the
  study presenting that risk, within 5 working days of that determination and within 15
  working days of first receipt of UADE notification as well as notify the applicable regulatory
  authorities.
- If the Sponsor confirms the reported event qualifies as a UADE, sponsor will notify the
  applicable regulatory authority(ies), all participating Investigators and reviewing IRBs/ECs
  within 10 working days of first receipt of UADE notification. Investigators are responsible
  for reviewing information received about UADEs.

UADEs will be recorded and followed until resolution or stabilization of the event or until the subject has exited the study.

#### 15.4 Sponsor Progress Reports

The Sponsor will submit progress reports with safety updates to the FDA, all participating Investigators, and all participating IRBs on at least an annual basis, as per federal regulations. These updates will be individualized for each institution and will include a summary of the study status, enrollment figures, any safety concerns, any outcomes, or recommendations from the Data Safety Monitoring Board (DSMB) as well as a listing of all adverse events reported.

#### 16 Statistics/Data Analyses

#### 16.1 Randomization

This is a randomized, controlled, open label study. Before the first subject is enrolled in the study, a randomization schedule will be generated by the study statistician and uploaded into an electronic database that can be accessed via computer. The schedule will be generated using a


Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


permuted block approach. Randomization will be performed at the conclusion of the index procedure, while the patient is on the table and the operator is able to visualize all access sites to verify eligibility. Since one of the primary endpoints of this study is time to ambulation, randomization will be done at the patient level to avoid the possibility of a patient receiving both MYNX CONTROL™ Venous VCD and manual compression. Randomization will be stratified by study center with a 2:1 randomization ratio for MYNX CONTROL™ Venous VCD vs. manual compression for access site closure. Roll-in patients will not be randomized. All roll-in patients will receive the MYNX CONTROL™ Venous VCD.

Any physician delegated as "Operator" on the Delegation of Authority log needs to have two (2) roll-in patients prior to randomizing any subject.

#### 16.2 Device Failures and Malfunctions

A device malfunction is considered a failure of a device to meet any of its performance specifications or otherwise perform as intended. Performance specifications include all claims made in the IFU/Clinical Protocol.

If a product malfunction occurs, the site must notify within 24 hours or one working day the Sponsor and/or enter details of the complication and its management in the respective CRF. If applicable, the malfunctioned product and any other materials used during the index procedure should be returned according to the Sponsor's instructions.

If a product malfunction occurs, detailed information on the product, circumstances of the malfunction as well as any complications and their management will be collected and reported.

Any patients randomized to the device arm who do not receive the MYNX CONTROL™ Venous VCD due to device malfunction would be treated with (converted to) manual compression, or much less likely – surgery – to close the access site. All device failure patients should be followed to 30 days and have a visual assessment of the access site(s) at that time. Such visual assessments are particularly important since patients experiencing device failures are more likely to have access site-related complications, and a complete and accurate evaluation of these patients is important to help ensure a rigorous IDE study.

#### 16.3 Analysis Population

Analyses for the safety and efficacy endpoints will be performed using the intent-to-treat (ITT) population. The ITT population will consist of all patients randomized in the study and will be analyzed in the group to which they were randomized regardless of the treatment actually received.

Supportive analyses for the safety and efficacy endpoints will be performed on the as-treated (AT) population and the per-protocol (PP) population. The AT population will consist of all randomized subjects, but they will be analyzed according to what device/treatment they actually received. The


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


PP population is a subset of the ITT population consisting of subjects that do not have any major protocol deviation that might affect the measurement of the primary endpoints.

#### 16.4 Statistical Hypotheses for Endpoints

Primary Effectiveness Endpoint- Primary efficacy will be measured using co-primary endpoints consisting of Time to Ambulation (TTA) and Time to Hemostasis (TTH) as defined below:

 Time to Ambulation (TTA)-Defined as elapsed time (in hours) between removal of the final VCD (device group) or of the final sheath (control group) and when subject stands and walks 20 feet without evidence of rebleeding from any femoral venous access site.

The null and alternative hypotheses of the primary effectiveness comparison for TTA are given below

Ho:  $\mu_{Mynx\ Control} \geq \mu_{manual\ compression}$ Ha:  $\mu_{Mynx\ Control} < \mu_{manual\ compression}$ 

Where  $\mu_x$  is the average time to ambulation for the specified group

 Time to Hemostasis (TTH)- Defined as elapsed time (in minutes) between removal of each VCD (device group) or of each sheath (control group) and first observed and confirmed venous hemostasis (per access site analysis)

The null and alternative hypotheses of the primary effectiveness comparison for TTH are given below:

Ho:  $\mu_{manual\ compression} - \mu_{Mynx\ Control} \le 5$ Ha:  $\mu_{manual\ compression} - \mu_{MynxControl} > 5$ 

Where  $\mu_{xx} \text{is}$  the mean time to hemostasis for the indicated group and 5 minutes is the superiority margin.

#### 16.5 Primary Safety Endpoint

The primary safety endpoint is defined as the rate of combined major venous access site closure- related complications through 30 days post procedure, attributed directly to VCD or manual compression without other likely cause.

- Access site-related bleeding requiring transfusion, surgical intervention, or rehospitalization
- Vascular injury requiring surgical repair
- Access site-related infection confirmed by culture and sensitivity, requiring intravenous antibiotics and/or extended hospitalization


100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




- New onset, permanent (i.e., persisting at 30-day follow-up) access site-related nerve injury
- New onset access site-related nerve injury requiring surgical repair
- Pulmonary embolism requiring surgical or endovascular intervention and/or resulting in death, to be confirmed by CT pulmonary angiography, lung ventilation/perfusion scan (VQ scan), or autopsy
- Pulmonary embolism not requiring surgical or endovascular intervention and/or not resulting in death, to be confirmed by CT pulmonary angiography or lung ventilation/perfusion scan (VQ scan)

The null and alternative hypotheses of the primary safety comparison are given below:

 $Ho: P_{Mynx\ Control} \geq P_{manual\ compression}$ 

 $Ha: P_{Mynx\ Control} < P_{manual\ compression}$ 

where  $P_X$  is the proportion limbs experiencing a major venous access site closure- related complications through 30 days post procedure and  $\delta$  is the non-inferiority window.

#### 16.6 Secondary Safety Endpoint

Rate of CEC adjudicated combined minor venous access site closure related complications within 30 days post\_procedure, attributed directly to VCD or manual compression without other likely cause.

- Pseudoaneurysm Treated with thrombin injection, fibrin adhesive injection, or ultrasound guided compression and documented by ultrasound
- Pseudoaneurysm Not requiring treatment
- · AV Fistula requiring treatment, documented by ultrasound
- · Arteriovenous fistula not requiring treatment, documented by ultrasound
- Access site related Hematoma > 6 cm documented by ultrasound
- Access site-related bleeding requiring > 30 min to achieve hemostasis
- Late access site-related bleeding (following hospital discharge eligibility)
- Transient loss of ipsilateral lower extremity pulse
- Ipsilateral deep vein thrombosis documented by ultrasound
- Transient access site-related nerve injury
- Access site-related vessel laceration
- Access site wound dehiscence
- Local access site infection confirmed by culture and sensitivity, treated with intramuscular or oral antibiotics – Minor
- Local access site inflammatory reaction Minor
- Allergic reaction
- Ecchymosis




100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


#### 16.7 Secondary Effectiveness Endpoints

- <u>Time to Discharge Eligibility</u>- defined as elapsed time (in hours) between removal of the final MYNX CONTROL™ Venous VCD (device group) or removal of the final sheath (control group) and when the subject is eligible for discharge from the institution based on the assessment of the attending physician.
- <u>Procedural Success</u>: attainment of final hemostasis at all venous access sites without major venous access site closure-related complications through 30 days.
- <u>Device Success</u>: ability to successfully deploy the MYNX CONTROL™ Venous VCD delivery system, deliver the polyethylene glycol hydrogel sealant, and achieve hemostasis (device group only).

#### 16.8 Sample Size Determination

In determining sample size for this study, it is necessary to take both TTA and TTH into account since the study is using both as co-primary endpoints. The total sample size for the study is determined to be 204 patients and is based on the following assumptions:

**TTA Assumptions** 

| Power | | 90% | | | |
|---|---|---|---|---|---|
| Alpha | | 1-sided 0.025 | | | |
| Allocation | | 2:1 VCD:MC | | | |
| VCD mean | | 3 hours <sup>78</sup> | | | |
| MC mean | | 6 hours | | | |
| Standard Devi | iation | 6 hours | | | |
| Attrition correction 5% | | | | | |
| Power | SD | | MC SS | VCD SS | Total SS |
| 90 | 6 | | 68 | 136 | 204 |

TTH Sample size justification: For the endpoint of time to hemostasis, a generalized linear mixed model will be used to compare the MYNX CONTROL™ Venous VCD device with manual compression (control). Initial estimates of the average time to hemostasis were taken from historical MYNX family devices and compared to manual compression. Previous MYNX family studies only studied one access site per subject within the femoral artery. The observed average time to hemostasis as well as the standard deviations of those measurements helped inform the design of this trial where the standard deviation would be used as an estimate of subject-to-subject variation. For the current study, it is assumed that each subject will have up to 4 access


ReliaSeal / P22-8301


sites in the femoral vein. These access sites will be closed with either the MYNX CONTROL™ Venous VCD device or manual compression. Only one method of closure will be used per subject. Time to hemostasis will be measured for each access site separately.

It is assumed that hemostasis times are log-normally distributed. Using previous study data, estimates of  $\mu$  and  $\sigma$  of the lognormal distribution were obtained and used in the calculation of sample size for this endpoint.

A generalized linear mixed model is used with the subject as a random effect. To adjust for the correlation in hemostasis time between the access sites within subject, it is assumed that the correlation structure is compound symmetric. The Type I error rate was set to a one-sided 0.025 (or equivalently, a two-sided 0.05 level) for the purposes of sample size calculation. A sample size of 150 patients (100 MYNX CONTROL<sup>TM</sup> Venous VCD and 50 manual compression) will provide approximately 95% power to detect a difference in hemostasis times of seven (7) minutes between MYNX CONTROL<sup>TM</sup> Venous VCD and manual compression. Note that these calculations were made in the log transformed space to assess power. Also, the variation between access sites within patients was estimated as approximately half of the variation observed between patients.

The specific model used is:

$$y_{ijk} = \mu + \tau_i + S_{j(i)} + e_{k(ij)}$$

where  $\tau_i$  is the treatment effect and  $S_{ij}$  is the random effect of subject within treatment.  $e_{ijk}$  is the unexplained variation in the model. Further, it is assumed that:

$$y_{ijk} \sim N(\mu_{ij}, \sigma^2)$$

$$S_{i(i)} \sim N(0, \sigma_S^2)$$

and

$$e_{k(ij)} \sim N(0, \sigma_e^2)$$

### **TTH Assumptions**

| Power | ~95% |
|----------------------|-----------------------------------------|
| Alpha | 1-sided 0.025 |
| Allocation | 2:1 VCD:MC |
| VCD mean | 6 |
| MC mean | 13 |
| Standard Deviation | Determined in the log transformed space |
| Attrition correction | 5% |




100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


| Total Sample Size | 150 patients |
|-------------------|--------------|

Sample Size for Primary Safety Endpoint: The primary safety endpoint of major venous access site closure-related complications through 30 days post-procedure, attributed directly to VCD or manual compression without other likely causes will be analyzed using a non-inferiority approach based on a generalized estimating equation (GEE) approach for logistic regression, using a working compound-symmetric covariance structure. This method would account for potential within subject correlation. We will perform the test at the one-sided 0.025 alpha level. For the purposes of sample size calculation, both groups are assumed to have a 1.5% major complication rate. The non-inferiority window has been established at 5 percentage points.

Within-subject correlation can affect the power of the study depending on the degree of correlation. However, the degree of correlation within-subject due to potentially multiple limbs is unknown and there is no robust and relevant data on which to base any associated assumption. Since this is unknown, sample size is conservatively calculated assuming only one limb per subject, or in other words, the number of subjects in the study assuming independence between subjects. Calculations for a two-sample test of binomial proportions for a Z test under a normal approximation show a sample size of 204 subjects should provide approximately 80% power for this endpoint. To the extent that some subjects will contribute multiple limbs to the actual analysis, the power would be higher than that from calculations based only on the number of independent subjects. Though missing data for the primary safety endpoint is unlikely, the additional data contributed by multiple limbs will help offset any power loss due to missing data.

Sample Size for Secondary Endpoint: Initial estimates for the secondary endpoint of time to discharge eligibility were obtained from the VASCADE MVP Venous Vascular Closure System (Cardiva Medical Inc.) Summary of Safety and Effectiveness Data. The average time to discharge eligibility for VASCADE was  $3.1 \pm 1.3$  hours and for manual compression it was  $6.5 \pm 1.9$  hours. For sample size calculation, the Type 1 error rate was set to 0.025. A sample size of 23 total subjects provides more than 95% power to demonstrate that the average time to discharge eligibility is significantly less for the MYNX CONTROL<sup>TM</sup> Venous group relative to manual compression.

The sample size for adequate power on the primary safety endpoint was the largest and will be used as the sample size for this trial.

#### 16.9 Statistical Analysis Methods

Except where otherwise specified, the following general principles apply to the planned statistical analyses. All descriptive statistical analyses will be performed using SAS version 9.4 or higher, unless otherwise noted (SAS Institute Inc., Cary, NC) or other widely accepted statistical or graphical software as required. Derived variables will be independently verified by an independent programmer / statistician. The program review will also include whether analyses conform to specifications of the Statistical Analysis Plan.


Protocol Clinical Clinical Study

Evaluation of Safety and Efficacy of Mynx Control Venous Vascular Closure Device 6F-12F (ReliaSeal)

Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


For categorical variables, the numerator, denominator, rate (%) and exact 95% CI will be calculated. For continuous variables, the median, mean, standard deviation, interquartile range, number of observations, minimum and maximum values, and 95% CI, as appropriate, will be presented.

For each parameter, the baseline value will be defined as the last non-missing value collected at the time closest to but before treatment with the investigational device.

All statistical tests will be performed at the two-sided 0.05 significance level, unless otherwise noted. Listings of patient data will be created for all study parameters.

16.9.1 Primary Analysis

# **Efficacy**

The primary efficacy endpoints will be analyzed separately.

The average time to ambulation in each treatment group will be compared using a standard T-test.

The average time to hemostasis will be compared to the treatment groups using a generalized linear mixed model where subject is considered a random effect with multiple access sites. The times to hemostasis in the manual compression group will be reduced by 5 minutes to account for the hypothesis that the time to hemostasis for the MYNX CONTROL™ Venous VCD is at least 5 minutes less than manual compression. The analysis will consist of testing the coefficient on the fixed effect for treatment group. If that coefficient is found to be significantly different from zero, then the direction will be evaluated to assure that the hemostasis time is reduced on average when using MYNX CONTROL ™ Venous VCD.

#### Safety

The safety analysis will be completed on a per-limb basis.

This endpoint will be analyzed using a GEE approach for a logistic regression model with a compound symmetric working covariance structure where occurrence of an AE is the binary response variable and treatment group is the only explanatory variable. Least square means for each treatment group and the risk difference between groups will be calculated along with the two-sided 95% confidence interval. The one-sided 97.5% confidence bound (equivalent to the appropriate bound from the two-sided 95% interval) will be compared to the non-inferiority window. If the upper bound is less than the non-inferiority window, then the two treatment groups will be considered non-inferior relative to the proportion of limbs experiencing a major venous access site closure-related complication.

As a supplementary analysis, a generalized linear mixed model will be used where subject will be entered into the model as a random effect and a compound symmetric correlation structure applied to those subjects contributing two limbs.


**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


#### **Trial Success**

This trial will be considered a success if both primary efficacy endpoints and the primary safety endpoint are achieved.

# 16.9.2 Secondary Safety Analysis

The secondary safety analysis of combined minor venous access site closure related complications within 30 days post-procedure, attributed directly to VCD or manual compression without other likely cause will be summarized on a per-limb basis. The proportion of limbs experiencing a minor closure related complication will be calculated for each treatment group along with 95% confidence intervals. The difference between the proportions will then be estimated along with a 95% confidence interval.

# 16.9.3 Secondary Efficacy Analyses

Time to Discharge Eligibility, defined as the elapsed time between removal of the final MYNX CONTROL™ Venous VCD (device group) or removal of the final sheath (control group), and when the subject is eligible for discharge from the institution (in hours) will be summarized on a perpatient basis.

Time to discharge eligibility is a powered secondary endpoint. The average time to discharge eligibility will be compared between the device and control groups at the 0.025 level of significance. The specific hypotheses being tested are:

 $Ho: \mu_{Mynx\ Control} \geq \mu_{manual\ compression}$ 

Ha:  $\mu_{Mynx\ Control} < \mu_{manual\ compression}$ 

where  $\mu_x$  is the average time to discharge eligibility for the specified group. A p-value for this one-sided test less than 0.025 will indicate that the time to discharge eligibility for the subjects using the MYNX CONTROL<sup>TM</sup> Venous Vascular Closure Device (VCD) was significantly less than for those where manual compression was used. The standard two group T-test will be used to make this comparison.

The difference between treatment groups in average time to discharge will also be estimated with 95% confidence intervals calculated using the T-distribution.

The following secondary endpoints are considered ad hoc analyses and are not powered.

Procedural Success defined as the attainment of final hemostasis at all venous access sites without major venous access site closure-related complications through 30 days will be summarized on a per access site basis and on a per-limb basis. Procedural success will be estimated for each treatment group separately with 95% confidence intervals followed by an


**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


estimate of the difference in procedural success between the treatment groups and a 95% confidence interval on the difference.

Device Success defined as the ability to deploy the VCD delivery system, deliver the polyethylene glycol hydrogel sealant, and achieve hemostasis will be summarized on a per access site basis for the device group only. The proportion of device successes will be estimated along with a 95% confidence interval.

# 16.9.4 Additional analysis

The type of major complication will also be compared on a per-limb basis. Frequency distributions for the type of complication will be constructed for each treatment group and the frequency distributions will be examined informally. This analysis is for information purposes only.

# 16.9.5 Analysis of Roll-in Subjects

The roll-in subjects will be summarized descriptively. No formal analysis will be done. Roll-in subjects will not be part of the main analysis population. Details can be found in the statistical analysis plan.

# 16.9.6 Study site poolability

Study site poolability for the primary endpoint of time to ambulation will be analyzed using a two-way analysis of variance (ANOVA) model. The first factor in this model will be treatment group and the second factor will be study site. The treatment group by study site interaction will also be added to the model. If the interaction term is not significant at the 0.15 level, then the study sites will be pooled for the analysis of this endpoint.

Study site poolability for the primary endpoint of time to hemostasis will be analyzed using the general linear mixed model outlined in section 16.8. To that model fixed effects for study site and treatment group by study site interaction will be added. If the interaction term is not significant at the 0.15 level, then the study sites will be pooled for the analysis of this endpoint.

Study site poolability for the safety endpoint will be analyzed on a per limb basis. A GEE logistic regression model with main effects of treatment group and study site along with an interaction term between those main effects will be fit to the data. If the interaction term is not significant at the 0.15 level, then the study sites will be pooled for the analysis of this endpoint.

# 16.9.7 Interim Analysis

An interim analysis in support of a CE Mark submission will be conducted to analyze initial subjects randomized to the device group only with respect to efficacy and safety. This interim analysis is not intended to support a decision to continue or to discontinue the trial, or to implement any modifications to trial procedures. To alleviate potential statistical and operational bias that may be introduced, the execution of the interim analysis shall be a completely confidential process to the study team. All sponsor staff, staff contracted by the sponsor, and investigator staff directly




involved in the conduct of the ongoing IDE trial will remain blind to the process and results of the analyses, with the exception of contracted resources involved in the execution of the interim analysis and submission of the results on behalf of the sponsor. Endpoints to be evaluated using descriptive statistics are as follows:

- Primary efficacy: Time to Ambulation and Time to Hemostasis.
- Secondary efficacy: Time to Discharge Eligibility, Procedure success, and Device Success.
  - Primary safety: rate of major complications related to the access site.
  - Secondary safety: rate of minor complications related to the access site.

This is a single-arm analysis, therefore subjects randomized to control arm will be excluded from the interim analysis. A sample size of 68 sequential subjects randomized to treatment arm will be collected for the interim analysis. A final clinical report will be prepared at the conclusion of the interim analysis by an agent of the sponsor who is independent from the conduct of the study. The report will be unblinded following the collection of the last patient's procedure data.

# 16.10 Sub-Group Analysis

A sub-group analysis will be completed for the primary safety and primary efficacy endpoints. This analysis is not powered and is strictly for information purposes. The sub-groups for this analysis are those subjects that contributed only 1 limb and those subjects that contributed 2 limbs. The same analysis outlined above for the primary safety and efficacy endpoints will be completed within each sub-group separately. Additional analyses to demonstrate the homogeneity of the treatment effect and homogeneity of the major complication rates are detailed in the SAP.

Major and minor complications will also be analyzed based on the number of access sites and sheath size, major and minor complications will be stratified by number of access sites per leg (1, 2, 3, or 4 sites), total number of access sites per patient (1, 2, 3, or 4 sites), and sheath size (small size vs. large size). Details are provided in the SAP.

A sub-group analysis will also be performed utilizing independent analysis of non-invasive duplex ultrasound (DUS) imaging in 72 subjects from both arms (48 device and 24 control) at the time of the procedure, pre-discharge and potentially again at the 30-day follow-up (only for those subjects that have documented evidence of access site complications at the discharge ultrasound). Specific investigational sites will be designated as ultrasound sites. These sites will include subjects in the ultrasound subset imaging until a total of 72 patients have been evaluated in both treatment arms. Ultrasound will be performed at the follow-up office visit only if a complication was detected at discharge. All sub-study sites will be instructed in performance of duplex ultrasonography of the femoral vascular structures. Images will be interpreted by:

NAMSA 4 World Trade Center


Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


150 Greenwich Street, 49<sup>th</sup> FL New York, NY 10007

At the time of the procedure, and at discharge, the proportion of subjects exhibiting a complication on DUS imaging will be calculated along with 95% confidence intervals constructed using the Clopper-Pearson method. For those subjects that required a DUS at the 30 day follow-up, the proportion of subjects still exhibiting a complication will be calculated along with a 95% confidence interval constructed using the Clopper-Pearson method.

#### 16.11 Missing Data

While all reasonable efforts will be made to obtain the data required to evaluate this endpoint, it is expected that some patients may not be able to provide data due to several reasons (loss to follow-up, study withdrawal, death). For all primary and secondary analyses, no imputation of missing data is planned. Patients who have ascertainment of status at a later out-of-window date (for example, patients who are known to be free of events past discharge eligibility but missed the discharge visit) are not considered missing as their status is known and their data will be used as noted previously. The primary endpoint rate will be calculated as the number of patients who had an event prior to the milestone visit divided by the number of evaluable patients who had sufficient follow up (e.g., at least discharge visit) plus any patients who had an event prior to the milestone visit. In other words, the denominator will be adjusted for missing follow up data.

A sensitivity analysis will be done to assess the impact of missing data on the conclusion of the primary analyses. Details of the analysis are provided in the SAP.

#### 16.12 Reporting

A final clinical summary will be developed for this study upon completion of all subject follow-up visits/database lock for the last required follow-up visit in the study.

This will be provided to the applicable regulatory authorities as well as all participating Investigators and Institutional Review Boards. Interim reports will also be developed and provided only as required.

# 17 Quality Control and Quality Assurance

# 17.1 Regulatory and Ethical Compliance

The Sponsor maintains a quality management system with written Standard Operating Procedures (SOP) to ensure that clinical studies are conducted, and data are generated, documented, and reported in compliance with the study protocol and the requirements of ICH E6 Good Clinical Practice, and the requirements of all applicable regulatory authorities. The staff at Cordis is trained regularly to ensure adherence to these SOPs.




100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


# 17.2 Data Quality Assurance

Study procedures to ensure the quality of all data collected and analyzed within this study include, but are not limited to, the following:

- Qualified Investigators, study sites and monitors will be selected.
- The investigational device was provided to Investigators/sites after being tested and released according to appropriate standards.
- Training will be provided to and documented for all Investigators and study personnel, which includes, but is not limited to, a review of the protocol, investigational product, CRFs, EDC system, GCP guidelines and study expectations. Training of Investigators will occur at the site initiation visit (prior to the start of any study-related activities), at any Investigator meetings and as necessary (e.g., when there are changes to the study team)
- Training will be provided to all study monitors on the study protocol, background/therapeutic area and GCP-conforming monitoring activities. Monitors will receive project-specific monitoring conventions and all forms needed to document the monitoring activity (e.g., forms for monitoring reports, investigational product accountability).
- The Sponsor and/or designee will conduct source document verification, as specified in the sponsor's monitoring plan by comparing original source documentation against the CRFs. Any discrepancies identified will be resolved with the Investigator, or designee, as appropriate.
- Appropriate edit checks incorporated within the EDC system and regular/periodic reviews
  of the data by Data Management will verify the completeness and accuracy of the data.
  Like the study monitor, Data Management will post queries to data points in need of further
  clarification and/or correction from sites (like the study monitor) and will keep the Sponsor
  informed of the status of queries and completeness of the study database.

### 17.3 Clinical Data

The case report form (CRF) for each subject is a record of their eligibility to enter the study, medical history, pre-procedure/baseline assessments, concomitant medications, all investigational product used during the index procedure, all procedural complications, and adverse events as well as data from discharge, all follow-up, and any unscheduled visits. It is the obligation of each Investigator (or designee) to ensure that all source documents (e.g., medical files, clinic charts, diagnostic films, nursing files), are available to support all data points collected within the CRF for every screened and/or enrolled subject. All information obtained during and between all protocol-required procedures needs to be clearly documented within the subject's source documentation and CRF.

Qualified site staff trained to the protocol, CRFs and EDC system will perform primary data collection and data entry into the CRFs in a timely manner following subject enrollment and/the completion of study-required assessments/follow-up visits. Data will be collected from patients' hospital charts, imaging films, and/or other medical records, which the Investigator is responsible to ensure are adequate to support all CRF entries. Corrections to CRFs will be performed by the


Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


Investigator or other authorized study site personnel. A record of study site personnel authorized to perform CRF data entry and/or corrections will be maintained by the site and provided to the Sponsor.

The Investigator must sign and date the specified section(s) within the CRF to confirm that s/he has reviewed the data and that the data are complete and accurate.

### 17.4 Monitoring

The Sponsor (and/or designee) will oversee the conduct and progress of the study at each investigational site. In addition to regular communications with the site, the Sponsor (and/or designee) will conduct interim monitoring visits (IMV) at periodic intervals to verify the following:

- The rights and well-being of the patients are protected
- The study is conducted according to International Council for Harmonization (ICH) and Good Clinical Practices (GCP) (ICH E6), the Declaration of Helsinki (1964) and all national, state, and local laws of the pertinent regulatory authorities
- The study is conducted in compliance with all requirements identified within the approved protocol/ amendment(s)
- The data reported in the CRFs/EDC system are accurate, complete, and verifiable from source documentation.

The study monitor will complete verification of the above primarily from review and assessment of regulatory documents, signed informed consent forms, accountability records and storage of investigational product and CRF/EDC system entries against all source documents. The monitor will also post and address queries within the EDC system and discuss the conduct of the study with the Investigator and study team. CRFs would need to be completed in a timely manner, within five (5) working days or one (1) week, to ensure availability for IMVs. Complete details regarding the monitoring procedures followed for the study are described in the study monitoring plan.

The Investigator must agree to provide study monitors with direct access to the office/clinic/facilities, medical records/source data/source documents for all enrolled patients, regulatory documents, and any/all other applicable study-related documents to enable the proper completion of IMVs.

Interim monitoring visits (IMVs) will be conducted throughout the course of this study according to the Sponsor's Monitoring Plan. Monitoring visit frequency at sites will be based on factors including, but not limited to, the rate and volume of enrollment, timing of completing follow-up visits and overall compliance.


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


#### 17.5 Protocol Modifications

#### 17.5.1 Protocol Amendments

Changes to the research covered by this protocol must be implemented through a formal protocol amendment. Change(s) to only logistical or administrative aspects of the study will be reflected in the study protocol if/when it is next amended to address any changes to the research. Protocol amendments may be initiated by the Sponsor or at the request of the Investigator. In either case, however, all protocol amendments must be approved by the Sponsor, signed, and dated by the Investigator and approved by the IRB prior to implementation.

#### 17.5.2 Protocol Deviations/Noncompliance

A protocol deviation is defined as a divergence from a specific element of the study protocol (e.g., missed assessment, visit out of window, violation of inclusion/exclusion criteria). Sites must comply with all requirements of the study protocol to control the number of protocol deviations to the extent possible. This does not include circumstances where necessary to eliminate an immediate hazard to study subjects (see section below) or that involve only logistical or administrative aspects of the study.

Protocol deviations for inability to perform office visits, exams or procedures due to COVID-19 pandemic should be completed and a notation of "COVID-19" in the CRF for each deviation.

The study monitor will verify the conduct of the study follows the currently approved protocol at each site and will identify any deviations from the protocol. The study monitor will also determine if there are any other issues of noncompliance (e.g., with IRB requirements, regulations from applicable regulatory authorities). If any protocol deviations or other areas of noncompliance are noted, the Investigator, site staff and/or study monitor will ensure corrective actions are implemented and evaluate the effectiveness of those corrective actions. Recurrence of noncompliance may require development of a formal corrective action plan that includes a suspension in enrollment and/or other actions. All protocol deviations and other issues of noncompliance at a site will be monitored closely by the Sponsor and/or designee(s) and will be reported to the applicable regulatory authorities and/or the IRB, as required.

### 17.5.3 Emergency Deviations

Emergency deviations are allowed <u>only</u> in cases where the change is necessary to eliminate an immediate apparent hazard and protect the life or physical well-being of a study subject. Such cases must be reported to the Sponsor/Medical Monitor and the IRB in writing within five (5) working days of the occurrence and will still be entered as protocol deviations in the CRF.

#### 17.6 Audits

The Sponsor and/or designee and the FDA may contact the participating institution to inform the Investigator of an upcoming audit and/or inspection, which may be routine or "for cause". In the


Protocol Clinical Clinical Study

Evaluation of Safety and Efficacy of Mynx Control Venous Vascular Closure Device 6F-12F (ReliaSeal)

Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


event the Investigator receives notification from FDA of an audit/inspection for this study, the Investigator should immediately notify the Sponsor. The Investigator must agree to provide direct access to the office/clinic/facilities, medical records/source documents for all enrolled patients, regulatory documents, and any/all other applicable study-related documents to all representatives of the Sponsor and/or designee and all regulatory authorities to enable proper completion of the audit/inspection.

# 17.7 Subject Confidentiality

Subject confidentiality will be maintained throughout the clinical study. A unique subject identification number will be assigned to every consented study subject, which will identify all data reported for that subject and ensure the data can be traced back to their source records. Subject identification will be created using a five-digit numeric value beginning with site number (XX) followed by subject numbers (YYY) such as 01-001.

Data relating to the study may be made available to all representatives of the Sponsor and/or designee and third parties (e.g., in the case of an audit performed by regulatory authorities) provided the data are treated confidentially and that the patient's privacy is guaranteed.

# 17.8 Institutional Review Board (IRB)

Prior to study initiation, the protocol, informed consent form and all other applicable study-related documents, including any written materials to be provided to patients, and any advertisement for patient recruitment (if applicable), must be submitted for review by a certified IRB. The IRB must be registered with the U.S. Department of Health and Human Services (HHS). Written approval or favorable opinion of these documents must be obtained and submitted to the Sponsor prior to screening and enrolling any patients and initiating any study-related activities.

The Investigator will prepare the draft informed consent form (ICF) and provide to the Sponsor and/or designee for approval prior to submission to the IRB. If the Sponsor requires any changes, a revised draft of the ICF incorporating these changes must be approved by the Sponsor prior to IRB submission. If the IRB requires additional changes, these must be reviewed and approved by the Sponsor prior to resubmission to the IRB. Copies of the final, IRB-approved ICF and all other IRB-approved study documents must be submitted to Sponsor or designee.

The Investigator or authorized designee will promptly report all changes in research activity and all unanticipated events/issues involving risks to human patients to the IRB. All Sponsor-approved amendments to the study protocol, ICF, etc. must be approved by the IRB prior to implementation. All other changes to research activities must be approved by the Sponsor and IRB prior to implementing, except when necessary to eliminate an immediate apparent hazard to the patient.

At least annually, or more frequently if required by IRB policy, the Investigator or authorized designee must submit a study progress report to their IRB to obtain continuing review approval for the study prior to the expiration of the most recent approval. Additionally, the Investigator must provide notification to their IRB, within three (3) months following the completion, termination, or


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


discontinuation of the study at the specific site and provide the acknowledgement letter from the IRB to the Sponsor.

For U.S. sites, IRBs must retain all study-related records for at least three (3) years following completion of the study, per the requirements of applicable regulatory authorities, or longer if required by local laws.

# 18 Record Keeping/Publication Policy

All required subject data must be recorded on CRFs provided by the Sponsor and/or designee for verification against subject source documents by the study monitor(s). A printout of the CRFs cannot be used as source documentation.

#### 18.1 Record Retention

All study records (e.g., correspondence, regulatory documents, CRFs and all source documents (informed consent forms, laboratory reports, progress notes, medical histories, physical and diagnostic findings, diagnoses, procedure/assessment dates and investigational product disposition records etc.) that support the CRFs) must be retained in the files of the responsible Investigator for a minimum of two (2) years from the latter of these two (2) dates, as communicated by the Sponsor, unless a longer retention period is required by the IRB or applicable local laws:

- the date on which the entire investigation is terminated or completed, or
- the date the records are no longer required to support a premarket approval (PMA) application

If the Investigator plans to archive or relocate/transfer the study records, (s)he must notify the Sponsor, in writing, of the transfer location, duration, and the procedure for accessing the study documentation. The Sponsor must approve of the planned archival or relocation/transfer, in writing, prior to its occurrence. All study records must be accessible upon request by the applicable regulatory authorities, the Sponsor and/or designee until destruction is possible.

If the Investigator retires, relocates, or for other reasons, withdraws from assuming primary responsibility for keeping the study records, written notice (transfer of obligation) must be submitted to the Sponsor and IRB indicating the name and address of the new custodian accepting primary responsibility.

For U.S. sites, IRBs must retain all study-related records for at least three (3) years following completion of the study, per the requirements of applicable regulatory authorities, or longer if required by local laws.

#### 18.2 Use of Information and Publications

This study will be registered in Clinicaltrials.gov, a publicly accessible database, through which the results of this study will also be reported. All information concerning the Sponsor (Cordis), MYNX CONTROL™ Venous Vascular Closure Device, patent application, manufacturing


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


processes, and scientific data supplied by the Sponsor to the Investigator and not previously published, is considered confidential and remains the sole property of the Sponsor. The Investigator understands the information developed in the clinical study will be used by the Sponsor in connection with a PMA application and thus may be disclosed as required to other Investigators or government regulatory authorities.

At the conclusion of the study, a manuscript may be prepared for publication of results across multiple study centers in a reputable scientific journal. The publication of the principal results from any single study center is not allowed until the preparation and publication of the multi-center results. Exceptions to this rule require prior approval of the Sponsor. The analysis of pre-specified and non-pre-specified endpoints will be performed by (the Sponsor/designated entity for data management/statistics). Secondary analyses as well as other proposed investigations will require the approval of the Sponsor. For purposes of timely abstract presentation and publication, secondary publications will be delegated to the appropriate principal authors.

# 19 Investigational Product Accountability

# 19.1 Study Investigational Product Accountability

The investigational product must be kept in a secure location with restricted access to authorized members of the study team and stored according to the conditions outlined in the Instructions for Use (IFU)/ Investigator Brochure (IB). The investigational product is intended solely for use by the Investigator or Sub-Investigator(s) and can only be used in clinical study patients. Investigational product-related study documentation to be maintained includes, but is not limited to, the following:

- Packing slips provided with each investigational product shipment (signed and dated)
- An up-to-date, complete, and accurate investigational product accountability log showing receipt, usage or implant and return or final disposition of all investigational product shipped to the site
- All other device accountability records including source documents and/or package labels of investigational product used in implanted patients, shipping labels, delivery confirmations, etc.
- Copies of investigational product malfunction and return forms (for sterile and opened/malfunctioned product)

All product on site labeled with "CAUTION Investigational device: Limited by Federal (or United States) law to investigational use.", regardless of whether used or opened and/or unused, will be inventoried and accounted for throughout the study. The Investigator and/or authorized designee will maintain adequate records of the receipt, use, and disposition of the investigational product as required by protocol and applicable country, local and federal regulations

Product on site will be inventoried and accounted for in the CRFs. At a minimum, the lot number, size (length and diameter) and use by date (UBD) of all products will be captured. All AEs, investigational product malfunctions and other product issues must also be recorded in the CRFs.


Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


# 19.2 Instructions for Return of Investigational Product

The Sponsor will provide instructions and ensure training to all sites on the re-package and return of investigational product, the appropriate form(s) that must be completed and the address(es) to which the product must be returned based on whether it is opened/unopened and unused, expired, damaged, mislabeled, a product complaint or malfunction has occurred, or study enrollment has been completed.

# 20 Committees

#### 20.1 Clinical Events Committee

The Clinical Events Committee (CEC) is responsible for the review and final adjudication of adverse events using source documents provided by sites to categorize clinical events and clinical endpoints in the study. The CEC will establish study-related guidelines for the requisite source data and the algorithm followed to classify a clinical event (according to the study definition). The Sponsor will review the definitions prior to the start of the adjudication process.

The CEC will consist of qualified physicians with the appropriate expertise for the type of investigational product or condition under study. The CEC is an independent body, functioning separately from the Sponsor, the investigational sites or anyone otherwise involved in the conduct of the study or the clinical care of study patients. Members will not have any scientific, financial, or other conflict of interest related to the Sponsor or the study Investigators. As appropriate, members of the CEC will be blinded to the primary results of the trial.

The CEC will be responsible for providing adjudication results and minutes of their meetings to the Sponsor for internal review.

The structure and function of the CEC will be documented in the CEC Charter.

### 20.2 Data and Safety Monitoring Board

The Data and Safety Monitoring Board (DSMB) is a body of professionals (primarily comprised of physicians, a biostatistician, and/or a medical ethicist) which reviews overall study data at intervals pre-determined before the start of the study and/or based on subject enrollment accrual and/or event accrual to assess progress and identify any safety concerns or other issues. The DSMB is independent of the Sponsor, the investigational sites or anyone otherwise involved in the conduct of the study. Members will not have any scientific, financial, or other conflict of interest related to the Sponsor or the study Investigators.

All serious adverse events, device-related complications/malfunctions and events related to the primary safety endpoint will be included in safety reports provided to the DSMB.


**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


The DSMB will be responsible for providing to the Sponsor, minutes of their meetings and any recommendations regarding early termination, suspension, or modifications to the study, if the safety and well-being of the patients is in jeopardy.

The structure and function of the DSMB will be documented in the DSMB Charter.

# 21 Early Termination or Suspension

The Sponsor, DSMB, IRBs, regulatory authorities or the Investigator may choose to temporarily suspend or prematurely terminate the study if the safety and well-being of the patients is in jeopardy.

The Sponsor reserves the right to temporarily suspend or prematurely terminate this study either at a single site, multiple sites or across all sites at any time for reasons including, but not limited to:

- Safety or ethical issues e.g., if in the opinion of the responsible investigator, the
  incidence and/or severity of adverse events in the study indicates a potential health
  hazard caused by treatment with the investigational product
- · Inaccurate or incomplete reporting of data
- Non-compliance
- Unsatisfactory enrollment with respect to quality or quantity
- Technical reasons (e.g., change in personnel)

If the Sponsor prematurely terminates or suspends the study, they will promptly notify the applicable Investigator(s)/institution(s) and the regulatory authority(ies) of the termination or suspension and the reason(s) for such, in accordance with applicable regulatory requirement(s). The applicable IRB(s)/EC(s) should also be informed and provided with the reason(s) for termination or suspension by the Sponsor or by the Investigator(s)/institution(s), in accordance with applicable regulatory requirement(s). Additionally, in the case of premature termination, the Sponsor will provide direction on the return of all unused investigational product and other study materials. In the case of a temporary suspension at a single site, multiple sites, or across all sites, the Sponsor will ensure all the necessary activities are performed before resuming the study, if approved to continue (e.g., benefit-risk reviewed and remain acceptable or revised).

If the Investigator terminates or suspends the study without prior agreement with the Sponsor, he/she will promptly provide all details to the institution, the Sponsor, and the IRB.

If the IRB terminates or suspends the study, the Investigator will promptly inform the Sponsor with written explanation.

In any case, the investigator(s)/institution(s) must arrange for any continued safety monitoring, treatment and/or follow-up of patients, unless it has been determined by the Investigator that the continued follow-up may jeopardize the rights, safety, and/or welfare of the subject.


Protocol Clinical Clinical Study

Evaluation of Safety and Efficacy of Mynx Control Venous Vascular Closure Device 6F-12F (ReliaSeal)

Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


Subject enrollment may be paused or terminated early if the Sponsor or DSMB determines that the potential benefits of the investigational product/procedure are unlikely to outweigh the risks. For example, if the probability of achieving the target primary endpoint falls below a certain threshold, the trial will be stopped or paused for re-evaluation.



100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


# Appendix A. Definitions

**Allergic reaction**: The hypersensitive response of the immune system of an allergic individual to a substance.

**Asymptomatic**: Without symptoms. For example, an asymptomatic infection is an infection with no symptoms.

Blood clot: Blood that has been converted from a liquid to a solid state. Also called a thrombus.

**Complication**: In medicine, an additional problem that arises following a procedure, treatment or illness and is secondary to it.

**Device related complication** - complication attributed to the device (e.g., graft migration, graft infection, etc.).

**Procedure-related complications** - complication not attributed to device but arises following the procedure (e.g., cardiac issue, renal insufficiency, etc.).

Death: All-cause mortality.

**Device deficiency:** Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. Includes malfunctions, use errors, and inadequate labelling.

**Device malfunction:** The failure of a device to meet any of its performance specifications or otherwise perform as intended. Performance specifications include all claims made in the IFU/IB.

**Dilation**: The process of enlargement, stretching, or expansion. The word "dilatation" means the same thing. Both come from the Latin "dilatare" meaning "to enlarge or expand."

**Inflammation**: A basic way in which the body reacts to infection, irritation or other injury, the key feature being redness, warmth, swelling and pain. Inflammation is now recognized as a type of nonspecific immune response.

Occlusion: A complete absence of flow within a blood vessel.

**Peripheral**: Situated away from the center, as opposed to centrally located.

Rupture: A break or tear in any organ or soft tissue

**Scan**: The data or image obtained from the examination of organs or regions of the body by gathering information with a sensing device.

**Stroke:** Any acute, new, persistent, documented neurological deficit ending in death or lasting greater than 24 hours and classified by a physician as a stroke.

Protocol Clinical Clinical Study

Evaluation of Safety and Efficacy of Mynx Control Venous Vascular Closure Device 6F-12F (ReliaSeal)

Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


**Thrombosis** – Formation of thrombus within a blood vessel leading to significant limitation of blood flow, requiring secondary intervention to restore blood flow (e.g., thrombolysis, thrombectomy, PTA)

**Ultrasound**: High-frequency sound waves used to bounce off tissues using special devices. The echoes are then converted into a picture called a sonogram.



100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301


# Appendix B. Acronyms and Abbreviation

| Acronym /<br>Abbreviation | Term |
|---|---|
| ADDIEVIATION | Activated platting time |
| AE | Activated clotting time Adverse event |
| AP | Anterior/Posterior |
| ARF w/ Dialysis | Acute Renal Failure with Dialysis |
| ARF w/o Dialysis | Acute Renal Failure without Dialysis |
| atm | Atmospheric pressure |
| AV | Arterial Venous |
| BID | Twice Daily |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| BUN | Blood urea nitrogen |
| CAD | Coronary Artery Disease |
| CAD | Carotid Artery Disease |
| CBC | Complete blood count |
| cc | cubic centimeter |
| CEC | Clinical Events Committee |
| CFA | Common Femoral Artery |
| CFR | Code of Federal Regulations |
| CHF | Coronary Heart Failure |
| CI | Confidence Interval |
| СК | Creatine kinase |
| CK-MB | Creatine kinase myocardial-band isoenzyme |
| cm | Centimeter |
| COPD | Chronic Obstructive Pulmonary Disease |
| CPK | Creatine Phosphokinase |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CSR | Clinical Study Report |
| CT | Computerized Axial Tomography Scan |
| CVA | Cerebrovascular accident |
| DIC | Disseminated Intravascular Coagulation |
| dl | deciliter |
| DM | Data Management |
| DSMB | Data and Safety Monitoring Board |
| DUS | Duplex Ultrasound |
| EC | Ethics Committee |
| eCRF | Electronic Case Report Form |
| EDC | |
| | Electronic Data Capture |
| Fr<br>GCP | French (sizing unit for devices) |
| | Good Clinical Practice |
| GGE | Generalized Estimating Equation |
| GI | Gastrointestinal |
| gm | Gram |
| HCT | Hematocrit |
| HGB | Hemoglobin |
| HHS | Health and Human Services (Department of) |
| HIPAA | Health Insurance Portability and Accountability Act |




100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301


| A avanym / | |
|---|---|
| Acronym / Abbreviation | Term |
| HR | Heart Rate |
| IB | Investigator Brochure |
| iCF | Informed Consent Form |
| ICH | International Council for Harmonization |
| ICU | Intensive Care Unit |
| IDE | Investigational Device Exemption |
| IFU | Instructions for Use |
| IMA | Inferior Mesenteric Artery |
| in | Inch |
| IRB | Institutional Review Board |
| ITT | Intent-to-treat |
| IV | Intravenous |
| IVRS | Interactive Voice Response System |
| IVUS | Intravascular ultrasound |
| LPO | Left Posterior Oblique |
| L/I | Liter |
| m/Mon | Month |
| MC | Manual Compression |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| MĬ | Myocardial infarction |
| mm | Millimeter |
| mmHg | Millimeters of mercury (unit of pressure) |
| MHLW | Ministry of Health, Labor and Welfare |
| NSTEMI | Non-ST segment Elevation Myocardial Infarction |
| NYHA | New York Heart Association |
| OR | Operation Room |
| PE | Physical Examination |
| PLT | Platelet |
| PMA | Premarket Approval |
| PMS | Post Marketing Surveillance study |
| PRN | As Required |
| RPO | Right Posterior Oblique |
| PRO | Patient-Reported Outcomes |
| PT | Prothrombin Time |
| PTA | Percutaneous transluminal angioplasty |
| PTT | Partial Thromboplastin Time |
| PVD | Peripheral Vascular Disease |
| QD | Once Daily |
| RBC | Red blood cell |
| RCT | Randomized Controlled Trial |
| RVD | Reference vessel diameter |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SMA | Superior Mesenteric Artery |
| SVS | Society for Vascular Surgery |
| TAA | Thoracic Aortic Aneurysm |
| TIA<br>TLR | Transient Ischemic Attack Target lesion(s) revascularization |
| ILIX | Target residin(s) revascularization |




100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301


| Acronym /<br>Abbreviation | Term |
|---------------------------|--------------------------------------------|
| TTA | Time to Ambulation |
| TTDE | Time to Discharge Eligibility |
| TTH | Time to Hemostasis |
| UADE | Unanticipated Adverse Device Effect |
| UBD | Use by date |
| ULN | Upper Limit of Normal |
| US/USA | United States/United States of America |
| USFDA | United States Food and Drug Administration |
| VCD | Vascular Closure Device |
| VO | Volume obstruction |
| WBC | White blood cell |
| WHO | World Health Organization |
| WNL | Within Normal Limit |

Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


# Appendix C. References

- 1. Moher D, Liberati A, Tetzlaff J, Altman DG. Preferred reporting items for systematic reviews and meta-analyses: the PRISMA statement. *PLoS medicine*. 2009;6(7):e1000097. 10.1371/journal.pmed.1000097
- 2. Baker NC, Escarcega RO, Lipinski MJ, Magalhaes MA, Koifman E, Kiramijyan S, et al. Active Versus Passive Anchoring Vascular Closure Devices Following Percutaneous Coronary Intervention: A Safety and Efficacy Comparative Analysis. *Journal of interventional cardiology*. 2016;29(1):108-12.10.1111/joic.12264
- 3. Fargen KM, Hoh BL, Mocco J. A prospective randomized single-blind trial of patient comfort following vessel closure: extravascular synthetic sealant closure provides less pain than a self-tightening suture vascular compression device. *Journal of neurointerventional surgery*. 2011;3(3):219-23.10.1136/jnis.2010.003988
- 4. Hutchings D, Hayat A, Karunakaran A, Malik N. Success, Safety, and Efficacy of the Mynx Femoral Closure Device in a Real-World Cohort: Single-Center Experience. *The Journal of invasive cardiology*.2016;28(3):104-8.
- 5. Noor S, Meyers S, Curl R. Successful reduction of surgeries secondary to arterial access site complications: a retrospective review at a single center with an extravascular closure device. *Vascular and endovascular surgery*. 2010;44(5):345-9. 10.1177/1538574410366760
- 6. Pruski MJ, Jr., Blachut AM, Konkolewska M, Janas A, Hrycek E, Buszman PP, et al. MynxGrip for Closure of Antegrade Puncture After Peripheral Interventions With Same-Day Discharge. *Vascular and endovascular surgery*. 2017;51(2):67-71. 10.1177/1538574416689424
- 7. Scheinert D, Sievert H, Turco MA, Schmidt A, Hauptmann KE, Mueller R, et al. The safety and efficacy of an extravascular, water-soluble sealant for vascular closure: initial clinical results for Mynx. *Catheterization and cardiovascular interventions: official journal of the Society for Cardiac Angiography & Interventions*. 2007;70(5):627-33. 10.1002/ccd.21353
- 8. Wong SC, Bachinsky W, Cambier P, Stoler R, Aji J, Rogers JH, et al. A randomized comparison of a novel bioabsorbable vascular closure device versus manual compression in the achievement of hemostasis after percutaneous femoral procedures: the ECLIPSE (Ensure's Vascular Closure Device Speeds Hemostasis Trial). *JACC Cardiovascular interventions*. 2009;2(8):785-93. 10.1016/j.jcin.2009.06.006
- 9. Sheth RA, Walker TG, Saad WE, Dariushnia SR, Ganguli S, Hogan MJ, et al. Quality improvement guidelines for vascular access and closure device use. *Journal of vascular and interventional radiology: JVIR*. 2014;25(1):73-84. 10.1016/j.jvir.2013.08.011
- 10. Rao SV, Stone GW. Arterial access and arteriotomy site closure devices. *Nature reviews Cardiology*. 2016;13(11):641-50. 10.1038/nrcardio.2016.133
- 11. Patel MR, Jneid H, Derdeyn CP, Klein LW, Levine GN, Lookstein RA, et al. Arteriotomy closure devices for cardiovascular procedures: a scientific statement from the American Heart Association. *Circulation*. 2010;122(18):1882-93. 10.1161/CIR.0b013e3181f9b345
- 12. Iannaccone M, Saint-Hilary G, Menardi D, Vadala P, Bernardi A, Bianco M, et al. Network metaanalysis of studies comparing closure devices for femoral access after percutaneous


100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




coronary intervention. *Journal of cardiovascular medicine (Hagerstown, Md)*. 2018.10.2459/jcm.00000000000000097

- 13. Kennedy SA, Rajan DK, Bassett P, Tan KT, Jaberi A, Mafeld S. Complication rates associated with antegrade use of vascular closure devices: a systematic review and pooled analysis. *Journal of vascular surgery*. 2020. 10.1016/j.jvs.2020.08.133
- 14. Schwartz BG, Burstein S, Economides C, Kloner RA, Shavelle DM, Mayeda GS. Review of vascular closure devices. *The Journal of invasive cardiology*. 2010;22(12):599-607.
- 15. Dahal K, Rijal J, Shahukhal R, Sharma S, Watti H, Azrin M, et al. Comparison of manual compression and vascular hemostasis devices after coronary angiography or percutaneous coronary intervention through femoral artery access: A meta-analysis of randomized controlled trials. *Cardiovascular revascularization medicine : including molecular interventions*. 2018;19(2):151-62.10.1016/j.carrev.2017.08.009
- 16. Noori VJ, Eldrup-Jørgensen J. A systematic review of vascular closure devices for femoral artery puncture sites. *Journal of vascular surgery*. 2018;68(3):887-99. 10.1016/j.jvs.2018.05.019
- 17. Vierhout BP, Pol RA, El Moumni M, Zeebregts CJ. Editor's Choice Arteriotomy Closure Devices in EVAR, TEVAR, and TAVR: A Systematic Review and Meta-analysis of Randomised Clinical Trials and Cohort Studies. *European journal of vascular and endovascular surgery: the official journal of the European Society for Vascular Surgery*. 2017;54(1):104-15. 10.1016/j.ejvs.2017.03.015
- 18. Rigattieri S, Sciahbasi A, Brilakis ES, Burzotta F, Rathore S, Pugliese FR, et al. Meta-Analysis of Radial Versus Femoral Artery Approach for Coronary Procedures in Patients With Previous Coronary Artery Bypass Grafting. *The American journal of cardiology*. 2016;117(8):1248-55.10.1016/j.amjcard.2016.01.016
- 19. Rigattieri S, Sciahbasi A, Ratib K, Alonzo A, Cox N, Chodor P, et al. Comparison Between Radial Approach and Femoral Approach With Vascular Closure Devices on the Occurrence of Access-Site Complications and Periprocedural Bleeding After Percutaneous Coronary Procedures: A Systematic Review and Meta-Analysis. *The Journal of invasive cardiology*. 2016;28(12):473-9.
- 20. Kiesz RS, Wiernek BK, Wiernek SL, Merritt C, Ybarra T, Iwanski A, et al. Cardiva Catalyst II vascular access management device in percutaneous diagnostic and interventional procedures with same-day discharge (Catalyst II trial). *Journal of endovascular therapy: an official journal of the International Society of Endovascular Specialists*. 2011;18(1):46-53. 10.1583/10-3237.1
- 21. Aksoy M, Becquemin JP, Desgranges P, Allaire E, Kobeiter H. The safety and efficacy of angioseal in therapeutic endovascular interventions. *European journal of vascular and endovascular surgery: the official journal of the European Society for Vascular Surgery*. 2006;32(1):90-3. 10.1016/j.ejvs.2005.12.014
- 22. Albert B, Davaine JM, Chaillet MP, Grimandi G, Guyomarch B, Azema L, et al. Clinical and economic evaluation of ambulatory endovascular treatment of peripheral arterial occlusive lesions. *Annals of vascular surgery*. 2014;28(1):137-43. 10.1016/j.avsg.2013.06.008


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


- 23. Alshehri AM, Elsharawy M. Comparison of Angioseal and Manual Compression in Patients Undergoing Transfemoral Coronary and Peripheral Vascular Interventional Procedures. *The International journal of angiology: official publication of the International College of Angiology, Inc.* 2015;24(2):133-6.10.1055/s-0035-1547449
- 24. Andrade PB, Mattos LA, Rinaldi FS, Bienert IC, Barbosa RA, Labrunie A, et al. Comparison of a vascular closure device versus the radial approach to reduce access site complications in non-ST-segment elevation acute coronary syndrome patients: The angio-seal versus the radial approach in acute coronary syndrome trial. *Catheterization and cardiovascular interventions:* official journal of the Society for Cardiac Angiography & Interventions. 2017;89(6):976-82. 10.1002/ccd.26689
- 25. Applegate RJ, Turi Z, Sachdev N, Ahmed A, Szyniszewski A, Foster M, et al. The Angio-Seal Evolution registry: outcomes of a novel automated Angio-Seal vascular closure device. *The Journal of invasive cardiology*. 2010;22(9):420-6.
- 26. Behan MW, Large JK, Patel NR, Lloyd GW, Sulke AN. A randomised controlled trial comparing the routine use of an Angio-Seal STS device strategy with conventional femoral haemostasis methods in a district general hospital. *International journal of clinical practice*. 2007;61(3):367-72. 10.1111/j.1742-1241.2006.01229.x
- 27. Brancheau D, Sarsam S, Assaad M, Zughaib M. Accelerated ambulation after vascular access closure device. *Therapeutic advances in cardiovascular disease*. 2018;12(5):141-4. 10.1177/1753944718756604
- 28. Burke MN, Hermiller J, Jaff MR. StarClose vascular closure system (VCS) is safe and effective in patients who ambulate early following successful femoral artery access closureresults from the RISE clinical trial. *Catheterization and cardiovascular interventions:* official journal of the Society for Cardiac Angiography & Interventions. 2012;80(1):45-52. 10.1002/ccd.23176
- 29. Chen CP, Huang HK, Hsia CH, Chang YM, Lin LS, Lee CL. Short-Term Safety and Efficacy of Femoral Vascular Closure after Percutaneous Coronary Intervention with Combination of the Boomerang(TM) Device and Intravenous Protamine Sulfate. *Acta Cardiologica Sinica*. 2013;29(6):531-8.
- 30. Chodor P, Kurek T, Kowalczuk A, Swierad M, Was T, Honisz G, et al. Radial vs femoral approach with StarClose clip placement for primary percutaneous coronary intervention in patients with STelevation myocardial infarction. RADIAMI II: a prospective, randomised, single centre trial. *Kardiologia polska*. 2011;69(8):763-71.
- 31. De Poli F, Leddet P, Couppie P, Daessle JM, Uhry S, Hanssen M. FemoSeal Evaluation Registry (FER). Prospective study of femoral arterial closure with a mechanical system on 100 patients who underwent angioplasty procedures. *Annales de cardiologie et d'angeiologie*. 2014;63(5):339-44.10.1016/j.ancard.2014.08.009
- 32. Deuling JH, Vermeulen RP, Anthonio RA, van den Heuvel AF, Jaarsma T, Jessurun G, et al. Closure of the femoral artery after cardiac catheterization: a comparison of Angio-Seal, StarClose, and manual compression. *Catheterization and cardiovascular interventions: official journal of the Society for Cardiac Angiography & Interventions*. 2008;71(4):518-23. 10.1002/ccd.21429


100606833 | Rev:4 Released: 19 May 2023

ReliaSeal / P22-8301




- 33. Fargen KM, Velat GJ, Lawson MF, Ritchie CA, Firment C, Hoh BL, et al. Occurrence of angiographic femoral artery complications after vascular closure with Mynx and AngioSeal. *Journal of neurointerventional surgery*. 2013;5(2):161-4. 10.1136/neurintsurg-2011-010217
- 34. Fastner C, Behnes M, Unsal M, El-Battrawy I, Ansari U, Mashayekhi K, et al. Clinical outcomes of femoral closure compared to radial compression devices following percutaneous coronary intervention: the FERARI study. *Heart and vessels*. 2017;32(5):520-30. 10.1007/s00380-016-0901-3
- 35. Fujihara M, Haramitsu Y, Ohshimo K, Yazu Y, Izumi E, Higashimori A, et al. Appropriate hemostasis by routine use of ultrasound echo-guided transfemoral access and vascular closure devices after lower extremity percutaneous revascularization. *Cardiovascular intervention and therapeutics*. 2017;32(3):233-40. 10.1007/s12928-016-0409-x
- 36. Goswami NJ, Smalling RG, Sinha S, Gammon RS, Ramaiah VG. Comparison of the boomerang wire vascular access management system versus manual compression alone during percutaneous diagnostic and interventional cardiovascular procedures: The boomerang wire vascular access management trial II. *Catheterization and cardiovascular interventions :* official journal of the Society for Cardiac Angiography & Interventions. 2016;87(1):75-81. 10.1002/ccd.25842
- 37. Heo YJ, Jeong HW, Baek JW, Lee SJ, Choo HJ, Jung HS, et al. Ultrasound Evaluation of Puncture Sites After Deployment of Two Different Types of Vascular Closure Devices: A Prospective Comparative Study. *Cardiovascular and interventional radiology*. 2018;41(11):1654-63. 10.1007/s00270-018-2056-3
- 38. Hermanides RS, Ottervanger JP, Dambrink JH, de Boer MJ, Hoorntje JC, Gosselink AT, et al. Closure device or manual compression in patients undergoing percutaneous coronary intervention: a randomized comparison. *The Journal of invasive cardiology*. 2010;22(12):562-6.
- 39. Hermiller JB, Leimbach W, Gammon R, Karas SP, Whitbourn RJ, Wong SC, et al. A prospective, randomized, pivotal trial of a novel extravascular collagen-based closure device compared to manual compression in diagnostic and interventional patients. *The Journal of invasive cardiology*. 2015;27(3):129-36.
- 40. Holm NR, Sindberg B, Schou M, Maeng M, Kaltoft A, Bottcher M, et al. Randomised comparison of manual compression and FemoSeal vascular closure device for closure after femoral artery access coronary angiography: the CLOSure dEvices Used in everyday Practice (CLOSE-UP) study. *EuroIntervention: journal of EuroPCR in collaboration with the Working Group on Interventional Cardiology of the European Society of Cardiology*. 2014;10(2):183-90. 10.4244/eijv10i2a31
- 41. Imam A, Carter RM, Phillips-Hughes J, Boardman P, Uberoi R. StarClose vascular closure device: prospective study on 222 deployments in an interventional radiology practice. *Cardiovascular and interventional radiology*. 2007;30(4):738-42. 10.1007/s00270-007-9079-5
- 42. Jensen J, Saleh N, Jensen U, Svane B, Jonsson A, Tornvall P. The inflammatory response to femoral arterial closure devices: a randomized comparison among FemoStop, AngioSeal, and Perclose. *Cardiovascular and interventional radiology*. 2008;31(4):751-5. 10.1007/s00270-008-9323-7


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


- 43. Jones LE, Yang KH, Feldtman RW, Uceda PV, Ferrara CA, Caruso JM, et al. Safety and Efficacy of Arterial Closure Devices in an Office-Based Angiosuite. *Annals of vascular surgery*. 2018;51:10-7.10.1016/j.avsg.2018.02.011
- 44. Kalsch HI, Eggebrecht H, Mayringer S, Konorza T, Sievers B, Sack S, et al. Randomized comparison of effects of suture-based and collagen-based vascular closure devices on post-procedural leg perfusion. *Clinical research in cardiology : official journal of the German Cardiac Society.* 2008;97(1):43-8. 10.1007/s00392-007-0575-z
- 45. Kara K, Kahlert P, Mahabadi AA, Plicht B, Lind AY, Longwitz D, et al. Comparison of collagen-based vascular closure devices in patients with vs. without severe peripheral artery disease. *Journal of endovascular therapy: an official journal of the International Society of Endovascular Specialists*. 2014;21(1):79-84. 10.1583/13-4401mr.1
- 46. Kara K, Mahabadi AA, Berg MH, Kahlert P, Longwitz D, Erbel R, et al. Utilization of collagen-based vascular closure devices in patients with severe peripheral artery disease. *The Journal of invasive cardiology*. 2013;25(1):19-22.
- 47. Ketterle J, Rittger H, Helmig I, Klinghammer L, Zimmermann S, Hohenforst-Schmidt W, et al. Comparison of Exo-Seal((R)) and Angio-Seal ((R)) for arterial puncture site closure: A randomized, multicenter, single-blind trial. *Herz.* 2015;40(5):809-16. 10.1007/s00059-015-4306-3
- 48. Klein-Wiele O, Baliota M, Kara K, Kaunicke M, Schafer H, Garbrecht M, et al. Safety and efficacy of clip-based vs. suture mediated vascular closure for femoral access hemostasis: A prospective randomized single center study comparing the StarClose and the ProGlide device. Catheterization and cardiovascular interventions: official journal of the Society for Cardiac Angiography & Interventions. 2018;91(3):402-7.10.1002/ccd.27116
- 49. Machnik R, Pieniążek P, Musiałek P, Przewłocki T, Tekieli Ł, Trystuła M, et al. Control of local haemostasis with the AngioSeal® vascular closure device in peripheral endovascular interventions via 6-9F femoral artery access. *Advances in Interventional Cardiology/Postępy w Kardiologii Interwencyjnej*. 2012;8(1):1-7. 10.5114/pwki.2012.27918
- 50. Manolis AS, Georgiopoulos G, Stalikas D, Koulouris S. Simplified swift and safe vascular closure device deployment without a local arteriogram: Single center experience in 2074 consecutive patients. *Indian heart journal*. 2016;68(4):529-38. 10.1016/j.ihj.2015.11.036
- 51. Martin JL, Pratsos A, Magargee E, Mayhew K, Pensyl C, Nunn M, et al. A randomized trial comparing compression, Perclose Proglide and Angio-Seal VIP for arterial closure following percutaneous coronary intervention: the CAP trial. *Catheterization and cardiovascular interventions: official journal of the Society for Cardiac Angiography & Interventions*. 2008;71(1):1-5. 10.1002/ccd.21333
- 52. Minko P, Katoh M, Graber S, Buecker A. Obesity: an independent risk factor for insufficient hemostasis using the AngioSeal vascular closure device after antegrade puncture. *Cardiovascular and interventional radiology.* 2012;35(4):775-8. 10.1007/s00270-011-0230-y
- 53. Rajan JE, Kannath SK, Sarma S, Kapilamoorthy TR. Prospective Evaluation of Factors Affecting the Safety and Efficacy of Perclose Proglide Vascular Closure Device in Neurovascular Interventions. *Neurology India*. 2019;67(5):1305-9. 10.4103/0028-3886.271252


Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


- 54. Rashid MN, Ahmed B, Straight F, Bradley JT, Gilbert K, Gogo PB, et al. Extravascular closure for patients with high-risk femoral anatomy. *The Journal of invasive cardiology*. 2008;20(7):328-32.
- 55. Rastan A, Sixt S, Schwarzwalder U, Schwarz T, Frank U, Burgelin K, et al. VIPER-2: a prospective, randomized single-center comparison of 2 different closure devices with a hemostatic wound dressing forclosure of femoral artery access sites. *Journal of endovascular therapy: an official journal of the International Society of Endovascular Specialists*. 2008;15(1):83-90. 10.1583/07-2253.1
- 56. Ratnam LA, Raja J, Munneke GJ, Morgan RA, Belli AM. Prospective nonrandomized trial of manual compression and Angio-Seal and Starclose arterial closure devices in common femoral punctures. *Cardiovascular and interventional radiology*. 2007;30(2):182-8. 10.1007/s00270-006-0226-1
- 57. Rittger H, Schmidt M, Breithardt OA, Mahnkopf C, Brachmann J, Sinha AM. Cardiorespiratory exercise testing early after the use of the Angio-Seal system for arterial puncture site closure after coronary angioplasty. *EuroIntervention: journal of EuroPCR in collaboration with the Working Group on Interventional Cardiology of the European Society of Cardiology*. 2011;7(2):242-7. 10.4244/eijv7i2a39
- 58. Sacherer M, Kolesnik E, von Lewinski F, Verheyen N, Brandner K, Wallner M, et al. Thermic sealing in femoral catheterization: First experience with the Secure Device. *Cardiology journal*. 2019;26(3):233-40. 10.5603/CJ.a2018.0035
- 59. Sato M, Matsumaru Y, Sakai N, Imamura H, Hirohata M, Takeuchi Y, et al. Usefulness of an accesssite hemostasis device in neuroendovascular treatment. *Acta neurochirurgica*. 2017;159(12):2331-5. 10.1007/s00701-017-3299-5
- 60. Sciahbasi A, Fischetti D, Picciolo A, Patrizi R, Sperduti I, Colonna G, et al. Transradial access compared with femoral puncture closure devices in percutaneous coronary procedures. *International journal of cardiology*. 2009;137(3):199-205. 10.1016/j.ijcard.2008.06.045
- 61. Sekhar A, Sutton BS, Raheja P, Mohsen A, Anggelis E, Anggelis CN, et al. Femoral arterial closure using ProGlide(R) is more efficacious and cost-effective when ambulating early following cardiac catheterization. *International journal of cardiology Heart & vasculature*. 2016;13:6-13. 10.1016/j.ijcha.2016.09.002
- 62. Spiliopoulos S, Kitrou P, Christeas N, Karnabatidis D. Starclose SE(R) hemostasis after 6F direct antegrade superficial femoral artery access distal to the femoral head for peripheral endovascular procedures in obese patients. *Diagnostic and interventional radiology (Ankara, Turkey)*. 2016;22(6):542-7. 10.5152/dir.2016.15614
- 63. Tavris DR, Wang Y, Jacobs S, Gallauresi B, Curtis J, Messenger J, et al. Bleeding and vascular complications at the femoral access site following percutaneous coronary intervention (PCI): an evaluation of hemostasis strategies. *The Journal of invasive cardiology*. 2012;24(7):328-34.
- 64. Tay EL, Co M, Tai BC, Lee YP, Low A, Lim YT, et al. Clinical experience of StarClose vascular closure device in patients with first and recurrent femoral punctures. *Journal of interventional cardiology*. 2008;21(1):67-73. 10.1111/j.1540-8183.2007.00291.x


Cordis

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


- 65. Teblick A, Vanderbruggen W, Vandendriessche T, Bosmans J, Haine SEF, Miljoen H, et al. Comparison of radial access versus femoral access with the use of a vascular closure device for the prevention of vascular complications and mortality after percutaneous coronary intervention. *Acta cardiologica*. 2018;73(3):241-7. 10.1080/00015385.2017.1363947
- 66. Veasey RA, Large JK, Silberbauer J, Paul G, Taggu W, Ellery S, et al. A randomised controlled trial comparing StarClose and AngioSeal vascular closure devices in a district general hospital--the SCOAST study. *International journal of clinical practice*. 2008;62(6):912-8. 10.1111/j.1742-1241.2008.01761.x
- 67. Wong HF, Lee CW, Chen YL, Wu YM, Weng HH, Wang YH, et al. Prospective comparison of angioseal versus manual compression for hemostasis after neurointerventional procedures under systemic heparinization. *AJNR American journal of neuroradiology*. 2013;34(2):397-401. 10.3174/ajnr.A3226
- 68. Wu PJ, Dai YT, Kao HL, Chang CH, Lou MF. Access site complications following transfemoral coronary procedures: comparison between traditional compression and angioseal vascular closure devices for haemostasis. *BMC cardiovascular disorders*. 2015;15:34. 10.1186/s12872-015-0022-4
- 69. Yeni H, Axel M, Ornek A, Butz T, Maagh P, Plehn G. Clinical and Subclinical Femoral Vascular Complications after Deployment of two Different Vascular Closure Devices or Manual Compression in the Setting of Coronary Intervention. *International journal of medical sciences*. 2016;13(4):255-9. 10.7150/ijms.14476
- 70. Tonolini M, Ierardi AM, Carrafiello G, Laganà D. Multidetector CT of iatrogenic and self-inflicted vascular lesions and infections at the groin. *Insights into imaging*. 2018;9(4):631-42. 10.1007/s13244-018-0613-6
- 71. Cox T, Blair L, Huntington C, Lincourt A, Sing R, Heniford BT. Systematic Review of Randomized Controlled Trials Comparing Manual Compression to Vascular Closure Devices for Diagnostic and Therapeutic Arterial Procedures. *Surgical technology international*. 2015;27:32-44.
- 72. Robertson L, Andras A, Colgan F, Jackson R. Vascular closure devices for femoral arterial puncture site haemostasis. *The Cochrane database of systematic reviews*. 2016;3:Cd009541. 10.1002/14651858.CD009541.pub2
- 73. Jiang J, Zou J, Ma H, Jiao Y, Yang H, Zhang X, et al. Network Meta-analysis of Randomized Trials on the Safety of Vascular Closure Devices for Femoral Arterial Puncture Site Haemostasis. *Scientific reports*. 2015;5:13761. 10.1038/srep13761
- 74. Resnic FS, Arora N, Matheny M, Reynolds MR. A cost-minimization analysis of the angio-seal vascular closure device following percutaneous coronary intervention. *The American journal of cardiology*. 2007;99(6):766-70. 10.1016/j.amjcard.2006.10.032
- 75. Ben-Dor I, Craig P, Torguson R, Rogers T, Buchanan KD, Pokharel S, et al. MynxGrip(R) vascular closure device versus manual compression for hemostasis of percutaneous transfemoral venous access closure: Results from a prospective multicenter randomized study. *Cardiovascular revascularization medicine : including molecular interventions*. 2018;19(4):418-22. 10.1016/j.carrev.2018.03.007


Cordis.

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


- 76. Mallow P, Belk K, Carver C, Almedhychy A, editors. Use of Vascular Closure Devices in the Hospital Setting for Percutaneous Coronary Procedures and Gender Differences of the Mynx® Vascular Closure Device: Results from a Hospital Claims Analysis. International Society for Pharmacoeconomics and Outcomes Research (ISPOR) 23rd Annual International Meeting; 2018; Baltimoare, MD, USA: Value in Health.
- 77. Boschewitz JM, Andersson M, Naehle CP, Schild HH, Wilhelm K, Meyer C. Retrospective evaluation of safety and effectiveness of the EXOSEAL vascular closure device for single vascular closure and closure after repeat puncture in diagnostic and interventional radiology: single-center experience. *Journal of vascular and interventional radiology : JVIR*. 2013;24(5):698-702. 10.1016/j.jvir.2013.02.014
- 78. Boschewitz JM, Pieper CC, Andersson M, Nadal J, Schild HH, Meyer C. Efficacy and time-to hemostasis of antegrade femoral access closure using the ExoSeal vascular closure device: a retrospective single-center study. *European journal of vascular and endovascular surgery: the official journal of the European Society for Vascular Surgery*. 2014;48(5):585-91. 10.1016/j.ejvs.2014.08.006
- 79. Grandhi R, Kanaan H, Shah A, Harrison G, Bonfield C, Jovin T, et al. Safety and efficacy of percutaneous femoral artery access followed by Mynx closure in cerebral neurovascular procedures: a single center analysis. *Journal of neurointerventional surgery*. 2014;6(6):445-50. 10.1136/neurintsurg-2013-010749
- 80. Grandhi R, Zhang X, Panczykowski D, Choi P, Hunnicutt CT, Jadhav AP, et al. Incidence of delayed angiographic femoral artery complications using the EXOSEAL vascular closure device. *Interventional neuroradiology : journal of peritherapeutic neuroradiology, surgical procedures and related neurosciences*. 2015;21(3):401-6. 10.1177/1591019915581776
- 81. Hackl G, Gary T, Belaj K, Hafner F, Rief P, Deutschmann H, et al. Exoseal for puncture site closure after antegrade procedures in peripheral arterial disease patients. *Diagnostic and interventional radiology (Ankara, Turkey)*. 2014;20(5):426-31. 10.5152/dir.2014.14002
- 82. Kara K, Mahabadi AA, Rothe H, Muller P, Kruger J, Neubauer H, et al. Safety and effectiveness of a novel vascular closure device: a prospective study of the ExoSeal compared to the Angio-Seal and ProGlide. *Journal of endovascular therapy: an official journal of the International Society of Endovascular Specialists*. 2014;21(6):822-8. 10.1583/14-4744mr.1
- 83. Maxien D, Behrends B, Eberhardt KM, Saam T, Thieme SF, Reiser MF, et al. Evaluation of the 6-F ExoSeal vascular closure device in antegrade femoral artery punctures. *Journal of endovascular therapy: an official journal of the International Society of Endovascular Specialists*. 2012;19(6):836-43. 10.1583/jevt-12-3922r.1
- 84. Pieper CC, Thomas D, Nadal J, Willinek WA, Schild HH, Meyer C. Patient Satisfaction After Femoral Arterial Access Site Closure Using the ExoSeal((R)) Vascular Closure Device Compared to Manual Compression: A Prospective Intra-individual Comparative Study. *Cardiovascular and interventional radiology*. 2016;39(1):21-7. 10.1007/s00270-015-1204-2
- 85. Rimon U, Khaitovich B, Yakubovich D, Bensaid P, Golan G, Silverberg D. The Use of ExoSeal Vascular Closure Device for Direct Antegrade Superficial Femoral Artery Puncture Site Hemostasis. *Cardiovascular and interventional radiology*. 2015;38(3):560-4. 10.1007/s00270-014-0984-0


**Cordis** 

100606833 | Rev:4

Released: 19 May 2023

ReliaSeal / P22-8301


86. Schelp V, Freitag-Wolf S, Hinzmann D, Bramlage P, Frey N, Frank D. Large-scale experience with an anchorless vascular closure device in a real-life clinical setting. *Clinical research in cardiology:* official journal of the German Cardiac Society. 2015;104(2):145-53. 10.1007/s00392-014-0766-3

87. Schmelter C, Liebl A, Poullos N, Ruppert V, Vorwerk D. Suitability of Exoseal vascular closure device for antegrade femoral artery puncture site closure. *Cardiovascular and interventional radiology*. 2013;36(3):659-68. 10.1007/s00270-012-0501-2
88. Moher D, Pham B, Lawson ML, Klassen TP. The inclusion of reports of randomised trials published in languages other than English in systematic reviews. *Health technology assessment (Winchester, England)*. 2003;7(41):1-90. 10.3310/hta7410